CLINICAL TRIAL: NCT02049138
Title: Phase 2 Study, Multicenter, Open-Label Extension (OLE) Study in Rheumatoid Arthritis Subjects Who Have Completed a Preceding Phase 2 Randomized Controlled Trial (RCT) With Upadacitinib (ABT-494)
Brief Title: An Open-label Extension Study Evaluating the Safety and Efficacy of Upadacitinib (ABT-494) in Adults With Rheumatoid Arthritis
Acronym: BALANCE-EXTEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-538; 2013-003530-33 (EudraCT Number)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Musculoskeletal Disease; Arthritis; Joint Diseases; Anti-inflammatory Agents; Antirheumatic agents
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — upadacitinib; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Upadacitinib (Experimental): Participants received treatment with upadacitinib for up to 312 weeks. The starting dose was 6 mg twice a day (BID). Participants who did not achieve a 20% improvement from RCT Baseline in both Tender Joint Count (TJC) and Swollen Joint Count (SJC) at Week 6 or Week 12 were up-titrated to 12 mg BID. From January 2017 participants were transitioned to a once-daily (QD) regimen of upadacitinib, either 15 mg QD (participants who were taking 6 mg BID) or 30 mg QD (participants taking 12 mg BID). Starting with Protocol Amendment 5 participants receiving 30 mg QD upadacitinib had the option to decrease the dose to 15 mg QD at the investigator's discretion.
  A subset of participants who opted-in to the vaccine substudy received a single-dose of 0.5 mL intramuscular injection of pneumococcal 13-valent conjugate vaccine (PCV-13).
  Interventions: Drug: Upadacitinib; Biological: Pneumococcal 13-valent conjugate vaccine (PCV-13)

INTERVENTIONS:
Drug: Upadacitinib — Tablet taken orally
  Other Names: ABT-494; RINVOQ®
Biological: Pneumococcal 13-valent conjugate vaccine (PCV-13) — Administered by intramuscular injection
  Other Names: Prevnar 13®

SUMMARY:
The primary objective of the study is to evaluate the long-term safety, tolerability, and efficacy of upadacitinib in adults with rheumatoid arthritis (RA) who have completed a preceding randomized controlled trial with upadacitinib.

DETAILED DESCRIPTION:
This is an open-label extension study to assess the long-term safety, tolerability, and efficacy of upadacitinib in adults with RA who have completed Study M13-550 (NCT01960855) or Study M13-537 (NCT02066389) Phase 2 randomized controlled trial (RCT) with upadacitinib.

All participants received treatment with 6 mg upadacitinib twice a day at the start of the study. Participants may have been up-titrated to 12 mg BID based on protocol-specified criteria. In Protocol Amendment 2 (January 2016) the study treatment was changed to a once daily (QD) formulation. Participants receiving 6 mg BID were transitioned to 15 mg QD and participants receiving 12 mg BID were transitioned to 30 mg QD dosing.

An optional 12-week vaccine sub-study was added in Protocol Amendment 3 (November 2017) to assess the impact of upadacitinib treatment (15 mg QD and 30 mg QD) with background methotrexate on immunological responses to pneumococcal 13-valent conjugate vaccine (PCV-13; Prevnar 13®) in RA patients. The vaccine substudy included 111 participants who were enrolled in the main study, the first participant was enrolled on 13 February 2018 and the the last participant completed the sub-study on 9 April 2020.

In Protocol Amendment 5 (December 2019), the protocol was revised to allow a decrease in upadacitinib dosing from 30 mg QD to 15 mg QD, as appropriate, based on investigator's medical decision or for safety/tolerability concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed Study M13-550 (NCT01960855) or Study M13-537 (NCT02066389) with upadacitinib (ABT-494) and did not develop any discontinuation criteria.
2. If the subject has evidence of new latent tuberculosis (TB) infection, the subject must initiate and complete a minimum of 2 weeks (or per local guidelines, whichever is longer) of an ongoing TB prophylaxis before continuing to receive study drug.
3. If female, subject must be postmenopausal, OR permanently surgically sterile, OR for women of childbearing potential practicing at least one protocol-specified method of birth control, that is effective from Study Day 1 through at least 30 days after the last dose of study drug.
4. Subjects must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures.

Substudy:

1. Must currently be enrolled in the main study.
2. Must have been receiving a stable dose of upadacitinib (either 15 mg QD or 30 mg QD) for a minimum of 4 weeks prior to the Vaccination visit.
3. Must have been on a stable dose of background methotrexate (no change in dose or frequency) for a minimum of 4 weeks prior to the Vaccination visit.
4. If subject is on corticosteroids, must remain on a stable dose of ≤ 10 mg/day of prednisone or equivalent corticosteroid therapy for at least 4 weeks after the vaccination visit.
5. Must meet the prescribing specifications as per local label requirements to receive Prevnar 13® vaccine.
6. Willing to receive Prevnar13® vaccine.

Exclusion Criteria:

1. Pregnant or breastfeeding female.
2. Ongoing infections at Week 0 that have not been successfully treated. Subjects with ongoing infections undergoing treatment may be enrolled but not dosed until the infection has been successfully treated.
3. Anticipated requirement or receipt of any live vaccine during study participation including up to 30 days after the last dose of study drug.
4. Laboratory values from the visit immediately prior to Baseline Visit (local requirements may apply) meeting the following criteria:

   * Serum aspartate transaminase (AST) or alanine transaminase (ALT) > 3.0 × upper limit of normal (ULN)
   * Estimated glomerular filtration rate by simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula < 40 mL/min/1.73m^2
   * Total white blood cell count (WBC) < 2,000/μL
   * Absolute neutrophil count (ANC) < 1,000/μL
   * Platelet count < 50,000/μL
   * Absolute lymphocytes count < 500/μL
   * Hemoglobin < 8 g/dL
5. Enrollment in another interventional clinical study while participating in this study.
6. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive study drug.

Substudy:

1. Receiving any conventional synthetic disease modifying antirheumatic drugs (csDMARDs) other than methotrexate
2. Receiving > 10 mg/day of prednisone or equivalent corticosteroid therapy.
3. Receipt of any steroid injection within 4 weeks prior to Vaccination visit.
4. History of severe allergic reaction (e.g., anaphylaxis) to any component of Prevnar 13®.
5. History of any documented pneumococcal infection within the last 6 months prior to the vaccination visit.
6. Receipt of any vaccine 4 weeks prior to the vaccination visit and/or anticipation of any vaccination for 4 weeks after the vaccination visit.
7. Receipt of any pneumococcal vaccine.
8. Subject is not suitable for the sub-study as per the Investigator's judgment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (124):
- United States (52):
  - Rheum Assoc of North Alabama /ID# 135926, Huntsville, Alabama
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 135902, Phoenix, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 135931, Phoenix, Arizona
  - C.V. Mehta MD, Med Corporation /ID# 124092, Hemet, California
  - Moores Cancer Center at UC San Diego /ID# 128747, La Jolla, California
  - Desert Medical Advances - Palm Desert /ID# 135911, Palm Desert, California
  - Orrin Troum, M.D. and Medical /ID# 135933, Santa Monica, California
  - Duplicate_Robin K. Dore MD, Inc /ID# 135906, Tustin, California
  - Inland Rheum Clin Trials Inc. /ID# 136716, Upland, California
  - Duplicate_Desert Valley Medical Group /ID# 135932, Victorville, California
  - Denver Arthritis Clinic /ID# 135901, Denver, Colorado
  - New England Research Associates, LLC /ID# 124085, Bridgeport, Connecticut
  - Arthritis & Rheumatic Disease Specialties /ID# 135910, Aventura, Florida
  - Rheumatology Associates of South Florida (RASF) - Clinical Research /ID# 124082, Boca Raton, Florida
  - Omega Research Maitland, LLC /ID# 124094, DeBary, Florida
  - University of Florida /ID# 124087, Jacksonville, Florida
  - Suncoast Research Group /ID# 137774, Miami, Florida
  - Omega Research Maitland, LLC /ID# 137398, Orlando, Florida
  - Millennium Research /ID# 135917, Ormond Beach, Florida
  - Arthritis Center, Inc. /ID# 124090, Palm Harbor, Florida
  - IRIS Research and Development, LLC /ID# 140362, Plantation, Florida
  - Lovelace Scientific Resources /ID# 128745, Venice, Florida
  - North Georgia Rheumatology Group /ID# 128746, Lawrenceville, Georgia
  - Kansas City Internal Medicine /ID# 135916, Overland Park, Kansas
  - PRN Professional Research Network of Kansas, LLC /ID# 124091, Wichita, Kansas
  - Klein and Associates MD - Hagerstown /ID# 124086, Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research /ID# 124077, Wheaton, Maryland
  - Clinical Pharmacology Study Group /ID# 124079, Worcester, Massachusetts
  - June DO, PC /ID# 124081, Lansing, Michigan
  - Summit Medical Group /ID# 124076, Clifton, New Jersey
  - Arthritis and Osteoporosis Associates /ID# 135907, Freehold, New Jersey
  - Arthritis Rheumatic and Back Disease Associates. P.A. /ID# 135913, Voorhees Township, New Jersey
  - Arthritis and Osteo Assoc /ID# 132280, Las Cruces, New Mexico
  - DJL Clinical Research, PLLC /ID# 131936, Charlotte, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Inc. /ID# 135921, Cincinnati, Ohio
  - STAT Research, Inc. /ID# 134906, Vandalia, Ohio
  - Health Research of Oklahoma /ID# 135904, Oklahoma City, Oklahoma
  - Duplicate_East Penn Rheumatology Assoc /ID# 135920, Bethlehem, Pennsylvania
  - Altoona Ctr Clinical Res /ID# 124089, Duncansville, Pennsylvania
  - Emkey Arthritis and Osteoporosis Clinic /ID# 135908, Wyomissing, Pennsylvania
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology /ID# 124080, Summerville, South Carolina
  - Dr. Ramesh Gupta /ID# 128744, Memphis, Tennessee
  - Austin Rheumatology Research /ID# 124083, Austin, Texas
  - Accurate Clinical Management /ID# 128751, Baytown, Texas
  - Accurate Clinical Management /ID# 128752, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 135905, Houston, Texas
  - Houston Institute for Clin Res /ID# 135912, Houston, Texas
  - Accurate Clinical Research /ID# 128753, Houston, Texas
  - Accurate Clinical Research /ID# 128754, Houston, Texas
  - SW Rheumatology Res. LLC /ID# 135927, Mesquite, Texas
  - Mountain State Clinical Research /ID# 124088, Clarksburg, West Virginia
  - Aurora Rheumatology and Immunotherapy Center /ID# 135922, Franklin, Wisconsin
- Belgium (2):
  - UCL Saint-Luc /ID# 139348, Woluwe-Saint-Lambert, Brussels Capital
  - ReumaClinic Genk-Hasselt /ID# 137775, Genk
- Bulgaria (7):
  - MHAT Trimontsium /ID# 135328, Plovdiv
  - Duplicate_MHAT Kaspela /ID# 136212, Plovdiv
  - UHMAT Palmed Plovdiv /ID# 135355, Plovdiv
  - UMHAT Sveti Ivan Rilski /ID# 135678, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 136210, Sofia
  - Diagnostic Consultative Center /ID# 136736, Sofia
  - Diagnostic consultative center Equita /ID# 136209, Varna
- Chile (2):
  - Corporacion de Beneficiencia Osorno /ID# 136189, Osorno, Los Lagos Region
  - Quantum Research /ID# 136188, Puerto Varas, Los Lagos Region
- Czechia (5):
  - Duplicate_Artroscan s.r.o. /ID# 139347, Ostrava
  - L.K.N. Arthrocentrum, s.r.o /ID# 128782, Petřkovice
  - Revmatologicky ustav v Praze /ID# 137937, Prague
  - Revmatologicka ambulance - MUDr. Zuzana Urbanova /ID# 137776, Prague
  - Revmatologie Bruntal, s.r.o /ID# 137782, Prostějov
- Hungary (5):
  - Qualiclinic Kft. /ID# 134170, Budapest, Pest County
  - Orszagos Reumatologiai es Fizioterapias Intezet /ID# 128785, Budapest
  - Szent Margit Szakrendelo /ID# 136676, Budapest
  - MAV Korhaz ess Rendelointezet /ID# 139971, Szolnok
  - Veszprem Megyei Csolnoky Ferenc Korhaz /ID# 128784, Veszprém
- Israel (2):
  - The Chaim Sheba Medical Center /ID# 139295, Ramat Gan, Tel Aviv
  - Barzilai Medical Center /ID# 140199, Ashkelon
- Latvia (3):
  - M & M Centrs LTD /ID# 132439, Ādaži
  - Arija's Ancane's Family Doctor Practice /ID# 132437, Baldone
  - Clinic ORTO /ID# 132438, Riga
- Mexico (3):
  - Clinstile, S.A. de C.V. /ID# 137075, Cuauhtémoc, Mexico City
  - Unidad de Investigacion de las Enfermedades Reumatologicas SA de CV /ID# 137307, Mexico City
  - Cliditer SA de CV /ID# 136876, Mexico City
- New Zealand (3):
  - Timaru Medical Specialists Ltd /ID# 131909, Timaru, Canterbury
  - Waikato Hospital /ID# 131908, Hamilton, Waikato Region
  - Porter Rheumatology Ltd /ID# 133983, Nelson
- Poland (14):
  - Prywatna Praktyka Lekarska /ID# 128837, Poznan, Greater Poland Voivodeship
  - Pratia MCM Krakow /ID# 134749, Krakow, Lesser Poland Voivodeship
  - Reum-Medica S.C. /ID# 128841, Wroclaw, Lower Silesian Voivodeship
  - Twoja Przychodnia Centrum Medyczne /ID# 128840, Nowa Sól, Lubusz Voivodeship
  - NZOZ Lecznica MAK-MED s.c. /ID# 128838, Nadarzyn, Masovian Voivodeship
  - Medicome sp. z o.o. /ID# 137397, Oswiecim, Masovian Voivodeship
  - NBR Polska /ID# 136208, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Amed Warszawa Zoliborz /ID# 128835, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia Warszawa /ID# 136650, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park w Warszawie /ID# 140198, Warsaw, Masovian Voivodeship
  - Gabinet Internistyczno-Reumatologiczny /ID# 135876, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 137362, Gdynia, Pomeranian Voivodeship
  - Ambulatorium Sp. z o.o /ID# 138074, Elblag, Warmian-Masurian Voivodeship
  - Duplicate_REUMED Filia nr 2 /ID# 128839, Lublin
- Puerto Rico (3):
  - Dr. Ramon L. Ortega-Colon, MD /ID# 128760, Carolina
  - GCM Medical Group PSC - Hato Rey /ID# 128759, San Juan
  - Mindful Medical Research /ID# 136211, San Juan
- Russia (3):
  - Kazan State Medical University /ID# 136734, Kazan', Tatarstan, Respublika
  - Tver Regional Clinical Hospital /ID# 137576, Tver', Tver Oblast
  - St. Petersburg Research Institute of Emergency Medicine n.а. I. I. Dzhanelidze /ID# 136652, Saint Petersburg
- Slovakia (2):
  - MEDMAN s.r.o. /ID# 136649, Martin
  - Poliklinika Senica n.o. /ID# 134728, Senica
- South Africa (2):
  - Dr MJ Prins /ID# 138540, Cape Town, Western Cape
  - Winelands Medical Research Centre /ID# 134669, Stellenbosch, Western Cape
- Spain (10):
  - Clinica Gaias /ID# 133868, Santiago de Compostela, A Coruna
  - Hospital General Universitario de Elche /ID# 128851, Elche, Alicante
  - Hospital Infanta Sofia /ID# 136653, San Sebastián de los Reyes, Madrid
  - Hospital Regional de Malaga /ID# 128847, Málaga, Malaga
  - Hospital Universitario A Coruna - CHUAC /ID# 128846, A Coruña
  - Hospital CIMA Sanitas /ID# 128849, Barcelona
  - Hospital Clinico Universitario San Carlos /ID# 128852, Madrid
  - Hospital Universitario Virgen Macarena /ID# 128853, Seville
  - Hospital QuironSalud Infanta Luisa /ID# 135689, Seville
  - Hospital Universitario Virgen de Valme /ID# 134668, Seville
- Ukraine (2):
  - NSC Strazhesko Ist Cardiology /ID# 137330, Kiev
  - Municipal Non-profit Institution Kyiv City Clinical Hospital No. 3 of the Exec /ID# 137334, Kyiv
- United Kingdom (4):
  - Warrington and Halton Hospitals NHS Foundation Trust /ID# 137514, Warrington, Cheshire West And Chester
  - Barts Health NHS Trust /ID# 135683, London, London, City of
  - West Suffolk Hospital /ID# 128858, Bury St Edmunds, Suffolk
  - Duplicate_Leeds Teaching Hospitals NHS Trust /ID# 141308, Leeds

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Baraliakos X, van der Heijde D, Sieper J, Inman RD, Kameda H, Li Y, Bu X, Shmagel A, Wung P, Song IH, Deodhar A. Efficacy and safety of upadacitinib in patients with ankylosing spondylitis refractory to biologic therapy: 1-year results from the open-label extension of a phase III study. Arthritis Res Ther. 2023 Sep 18;25(1):172. doi: 10.1186/s13075-023-03128-1. PMID 37723577
- [Derived] Kivitz A, Wells AF, Vargas JI, Baraf HSB, Rischmueller M, Klaff J, Khan N, Li Y, Carter K, Friedman A, Durez P. Long-Term Efficacy and Safety of Upadacitinib in Patients with Rheumatoid Arthritis: Final Results from the BALANCE-EXTEND Open-Label Extension Study. Rheumatol Ther. 2023 Aug;10(4):901-915. doi: 10.1007/s40744-023-00557-x. Epub 2023 May 18. PMID 37199884
- [Derived] Winthrop K, Vargas JI, Drescher E, Garcia C, Friedman A, Hendrickson B, Li Y, Klaff J, Kivitz A. Evaluation of response to 13-valent conjugated pneumococcal vaccination in patients with rheumatoid arthritis receiving upadacitinib: results from a phase 2 open-label extension study. RMD Open. 2022 Mar;8(1):e002110. doi: 10.1136/rmdopen-2021-002110. PMID 35246470
- See also: Related Info. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have completed a preceding rheumatoid arthritis (RA) upadacitinib randomized controlled trial (RCT), Study M13-550 (NCT01960855) or Study M13-537 (NCT02066389) to be enrolled in this long-term extension study.
  Participants were enrolled at 113 study sites located in 17 countries (Belgium, Bulgaria, Chile, Czechia, Hungary, Israel, Latvia, Mexico, New Zealand, Poland, Russian Federation, Slovakia, South Africa, Spain, United Kingdom, Ukraine, and United States/Puerto Rico).
Pre-assignment Details: Participants were assigned to upadacitinib 6 mg twice-daily up to 30 days following the Last Visit (Week 12) of the preceding RCT. Participants may have been up-titrated to 12 mg BID and subsequently down-titrated per protocol-specified criteria. Efficacy results are reported by treatment sequence for each participant. Adverse event data are reported according to treatment received at the time of the event.
  Participants may have enrolled in a vaccine substudy during the main study.
Groups:
- Upadacitinib Never Titrated: Participants received treatment with upadacitinib for up to 312 weeks. The starting dose was 6 mg twice a day (BID). From January 2017 participants were transitioned to a once-daily (QD) dose of 15 mg upadacitinib and remained on this dose throughout the study.
  A subset of participants who opted-in to the vaccine substudy received a single-dose of 0.5 mL intramuscular injection of pneumococcal 13-valent conjugate vaccine (PCV-13).
- Upadacitinib Titrated Up and Not Down: Participants received treatment with upadacitinib for up to 312 weeks. The starting dose was 6 mg BID. Participants who did not achieve protocol-specified improvement criteria at Week 6 or at any visits thereafter were up-titrated to upadacitinib 12 mg BID. From January 2017 participants were transitioned to a once-daily dose of 30 mg upadacitinib and remained on this dose throughout the study.
  A subset of participants who opted-in to the vaccine substudy received a single-dose of 0.5 mL intramuscular injection of pneumococcal 13-valent conjugate vaccine (PCV-13).
- Upadacitinib Titrated Up and Down: Participants received treatment with upadacitinib for up to 312 weeks. The starting dose was 6 mg BID. Participants who did not achieve protocol-specified improvement criteria at Week 6 or at any visits thereafter were up-titrated to upadacitinib 12 mg BID. From January 2017 participants were transitioned to once-daily dose of 30 mg upadacitinib. The upadacitinib dose was decreased back to 6 mg BID (or 15 mg QD from January 2017) per Investigator's judgment or safety and/or tolerability concerns.
  A subset of participants who opted-in to the vaccine substudy received a single-dose of 0.5 mL intramuscular injection of pneumococcal 13-valent conjugate vaccine (PCV-13).
Period: Overall Study
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Started | 306 | 149 | 38
Enrolled in Vaccine Sub-study | 76 | 24 | 11
Completed | 142 | 51 | 30
Not Completed | 164 | 98 | 8
Not completed — Adverse Event | 46 | 25 | 1
Not completed — Withdrawal by Subject | 57 | 21 | 5
Not completed — Lost to Follow-up | 18 | 5 | 1
Not completed — Lack of Efficacy | 10 | 26 | 1
Not completed — Non-Compliance | 15 | 6 | 0
Not completed — Required Alternative / Prohibited Therapy | 1 | 1 | 0
Not completed — Coronavirus Disease-2019 (COVID-19) Infection | 1 | 0 | 0
Not completed — COVID-19 Logistical Restrictions | 1 | 0 | 0
Not completed — Other | 15 | 13 | 0
Not completed — Missing | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The open-label treated population consisted of all participants who had received at least one dose of open-label study medication.
  Baseline data are from the Baseline of the preceding RCT study (M13-550 or M13-537).
Groups:
- Upadacitinib Never Titrated: Participants received treatment with upadacitinib for up to 312 weeks. The starting dose was 6 mg twice a day (BID). From January 2017 participants were transitioned to once-daily (QD) dose of 15 mg upadacitinib.
- Upadacitinib Titrated Up and Not Down: Participants received treatment with upadacitinib for up to 312 weeks. The starting dose was 6 mg BID. Participants who did not achieve protocol-specified improvement criteria at Week 6 or at any visits thereafter were up-titrated to upadacitinib 12 mg BID. From January 2017 participants were transitioned to once-daily dose of 30 mg upadacitinib.
- Upadacitinib Titrated Up and Down: Participants received treatment with upadacitinib for up to 312 weeks. The starting dose was 6 mg BID. Participants who did not achieve protocol-specified improvement criteria at Week 6 or at any visits thereafter were up-titrated to upadacitinib 12 mg BID. From January 2017 participants were transitioned to once-daily dose of 30 mg upadacitinib. The upadacitinib dose was decreased back to 6 mg BID (or 15 mg QD from January 2017) per Investigator's judgment or safety and/or tolerability concerns.
- Total: Total of all reporting groups
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down | Total
Number analyzed (Participants) | 306 | 149 | 38 | 493
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (12.62) | 56.0 (12.56) | 53.7 (8.54) | 55.7 (12.33)
Age, Customized [Count of Participants; unit: Participants]
  < 45 years | 56 | 30 | 5 | 91
  45 - < 65 years | 174 | 76 | 28 | 278
  ≥ 65 years | 76 | 43 | 5 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 117 | 29 | 392
  Male | 60 | 32 | 9 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 40 | 7 | 123
  Not Hispanic or Latino | 230 | 109 | 31 | 370
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 293 | 132 | 37 | 462
  Black or African American | 9 | 12 | 1 | 22
  Asian | 1 | 2 | 0 | 3
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Multiple | 2 | 3 | 0 | 5
Region [Count of Participants; unit: Participants]
  Western Europe | 27 | 13 | 5 | 45
  Eastern Europe | 144 | 46 | 19 | 209
  North America | 90 | 78 | 10 | 178
  South/Central America | 42 | 5 | 3 | 50
  Other | 3 | 7 | 1 | 11
Duration of RA [Mean (Standard Deviation); unit: years] | 9.34 (8.73) | 9.61 (8.36) | 7.66 (6.54) | 9.29 (8.47)
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  joints | 25.8 (14.49) | 30.4 (15.90) | 31.3 (15.67) | 27.6 (15.17)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  joints | 16.7 (10.45) | 18.8 (12.03) | 19.3 (9.53) | 17.5 (10.92)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: score on a scale] — The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a visual analog scale (VAS) from 0 to 100 mm, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 298 | 147 | 38 | 483
    (all) | 64.4 (15.82) | 65.6 (15.41) | 65.0 (15.41) | 64.8 (15.64)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: score on a scale] — The participant was asked to rate their current RA disease activity over the past 24 hours on a 100 mm VAS, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 305 | 146 | 37 | 488
    (all) | 62.4 (20.78) | 67.4 (20.52) | 66.5 (16.48) | 64.2 (20.51)
Patient's Global Assessment of Pain [Mean (Standard Deviation); unit: score on a scale] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale from 0 to 100 mm. A score of 0 mm indicates "no pain" and a score of 100 mm indicates "worst possible pain." Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 305 | 146 | 37 | 488
    (all) | 63.8 (19.73) | 67.2 (19.64) | 66.5 (13.13) | 65.0 (19.32)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: score on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 304 | 146 | 37 | 487
    (all) | 1.4811 (0.6848) | 1.6036 (0.6215) | 1.5304 (0.4969) | 1.5216 (0.6550)
High-sensitivity reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 12.8968 (17.8329) | 14.9212 (20.1890) | 17.1232 (28.1184) | 13.8344 (19.5179)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response Over Time
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline (of the preceding RCT study) and Weeks 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, and 312
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Groups:
- Upadacitinib Never Titrated: Participants received treatment with upadacitinib for up to 312 weeks. The starting dose was 6 mg twice a day (BID). From January 2017 participants were transitioned to once-daily dose of 15 mg upadacitinib.
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 277 | 143 | 36
  Week 6 | 87.7 | 73.4 | 77.8
  Week 12: number analyzed (Participants) | 273 | 141 | 37
  Week 12 | 89.0 | 73.8 | 75.7
  Week 24: number analyzed (Participants) | 256 | 131 | 35
  Week 24 | 91.8 | 73.3 | 88.6
  Week 36: number analyzed (Participants) | 246 | 125 | 35
  Week 36 | 90.2 | 83.2 | 82.9
  Week 48: number analyzed (Participants) | 229 | 117 | 34
  Week 48 | 90.0 | 82.1 | 88.2
  Week 60: number analyzed (Participants) | 217 | 105 | 35
  Week 60 | 95.4 | 83.8 | 85.7
  Week 72: number analyzed (Participants) | 199 | 101 | 32
  Week 72 | 93.0 | 84.2 | 90.6
  Week 84: number analyzed (Participants) | 203 | 97 | 32
  Week 84 | 94.6 | 76.3 | 96.9
  Week 96: number analyzed (Participants) | 204 | 93 | 33
  Week 96 | 92.2 | 86.0 | 90.9
  Week 108: number analyzed (Participants) | 194 | 91 | 33
  Week 108 | 94.8 | 85.7 | 87.9
  Week 120: number analyzed (Participants) | 186 | 86 | 29
  Week 120 | 96.2 | 89.5 | 96.6
  Week 132: number analyzed (Participants) | 181 | 80 | 30
  Week 132 | 93.9 | 87.5 | 96.7
  Week 144: number analyzed (Participants) | 178 | 75 | 27
  Week 144 | 94.9 | 88.0 | 88.9
  Week 156: number analyzed (Participants) | 176 | 73 | 27
  Week 156 | 92.0 | 87.7 | 92.6
  Week 168: number analyzed (Participants) | 172 | 71 | 29
  Week 168 | 91.9 | 88.7 | 82.8
  Week 180: number analyzed (Participants) | 179 | 67 | 29
  Week 180 | 93.9 | 79.1 | 86.2
  Week 192: number analyzed (Participants) | 168 | 70 | 28
  Week 192 | 93.5 | 87.1 | 92.9
  Week 204: number analyzed (Participants) | 166 | 69 | 29
  Week 204 | 94.0 | 81.2 | 86.2
  Week 216: number analyzed (Participants) | 160 | 64 | 27
  Week 216 | 92.5 | 85.9 | 85.2
  Week 228: number analyzed (Participants) | 149 | 55 | 28
  Week 228 | 96.0 | 83.6 | 92.9
  Week 240: number analyzed (Participants) | 153 | 61 | 28
  Week 240 | 92.8 | 85.2 | 89.3
  Week 252: number analyzed (Participants) | 149 | 58 | 30
  Week 252 | 94.0 | 87.9 | 86.7
  Week 264: number analyzed (Participants) | 135 | 54 | 28
  Week 264 | 93.3 | 81.5 | 89.3
  Week 276: number analyzed (Participants) | 128 | 52 | 27
  Week 276 | 93.8 | 84.6 | 81.5
  Week 288: number analyzed (Participants) | 133 | 50 | 27
  Week 288 | 94.7 | 88.0 | 88.9
  Week 300: number analyzed (Participants) | 125 | 50 | 23
  Week 300 | 94.4 | 82.0 | 87.0
  Week 312: number analyzed (Participants) | 129 | 49 | 26
  Week 312 | 92.2 | 87.8 | 88.5

2. Primary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response Over Time
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: as for outcome 1
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 275 | 144 | 35
  Week 6 | 63.6 | 37.5 | 48.6
  Week 12: number analyzed (Participants) | 275 | 141 | 35
  Week 12 | 73.5 | 41.8 | 45.7
  Week 24: number analyzed (Participants) | 251 | 131 | 35
  Week 24 | 75.7 | 49.6 | 60.0
  Week 36: number analyzed (Participants) | 245 | 126 | 34
  Week 36 | 73.5 | 51.6 | 55.9
  Week 48: number analyzed (Participants) | 229 | 116 | 36
  Week 48 | 74.2 | 50.0 | 55.6
  Week 60: number analyzed (Participants) | 213 | 108 | 35
  Week 60 | 79.8 | 52.8 | 65.7
  Week 72: number analyzed (Participants) | 201 | 102 | 33
  Week 72 | 77.1 | 49.0 | 63.6
  Week 84: number analyzed (Participants) | 203 | 95 | 33
  Week 84 | 78.8 | 55.8 | 75.8
  Week 96: number analyzed (Participants) | 202 | 93 | 33
  Week 96 | 74.8 | 53.8 | 63.6
  Week 108: number analyzed (Participants) | 194 | 93 | 34
  Week 108 | 79.4 | 54.8 | 58.8
  Week 120: number analyzed (Participants) | 187 | 88 | 29
  Week 120 | 80.7 | 58.0 | 72.4
  Week 132: number analyzed (Participants) | 178 | 80 | 29
  Week 132 | 79.2 | 56.3 | 69.0
  Week 144: number analyzed (Participants) | 178 | 73 | 28
  Week 144 | 76.4 | 65.8 | 60.7
  Week 156: number analyzed (Participants) | 176 | 71 | 26
  Week 156 | 79.5 | 63.4 | 76.9
  Week 168: number analyzed (Participants) | 173 | 72 | 29
  Week 168 | 79.2 | 61.1 | 75.9
  Week 180: number analyzed (Participants) | 178 | 70 | 29
  Week 180 | 80.9 | 64.3 | 65.5
  Week 192: number analyzed (Participants) | 166 | 69 | 26
  Week 192 | 80.7 | 59.4 | 76.9
  Week 204: number analyzed (Participants) | 163 | 69 | 29
  Week 204 | 82.2 | 59.4 | 79.3
  Week 216: number analyzed (Participants) | 158 | 63 | 27
  Week 216 | 76.6 | 55.6 | 66.7
  Week 228: number analyzed (Participants) | 149 | 55 | 28
  Week 228 | 79.2 | 58.2 | 67.9
  Week 240: number analyzed (Participants) | 152 | 61 | 28
  Week 240 | 79.6 | 63.9 | 71.4
  Week 252: number analyzed (Participants) | 148 | 58 | 30
  Week 252 | 83.8 | 55.2 | 76.7
  Week 264: number analyzed (Participants) | 133 | 55 | 28
  Week 264 | 79.7 | 60.0 | 75.0
  Week 276: number analyzed (Participants) | 129 | 51 | 27
  Week 276 | 84.5 | 52.9 | 66.7
  Week 288: number analyzed (Participants) | 135 | 51 | 26
  Week 288 | 82.2 | 58.8 | 61.5
  Week 300: number analyzed (Participants) | 127 | 49 | 23
  Week 300 | 75.6 | 61.2 | 56.5
  Week 312: number analyzed (Participants) | 127 | 49 | 26
  Week 312 | 84.3 | 69.4 | 69.2

3. Primary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response Over Time
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: as for outcome 1
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 273 | 146 | 37
  Week 6 | 38.8 | 15.1 | 21.6
  Week 12: number analyzed (Participants) | 274 | 144 | 37
  Week 12 | 47.1 | 18.1 | 24.3
  Week 24: number analyzed (Participants) | 253 | 134 | 35
  Week 24 | 45.5 | 27.6 | 37.1
  Week 36: number analyzed (Participants) | 243 | 127 | 35
  Week 36 | 49.0 | 28.3 | 34.3
  Week 48: number analyzed (Participants) | 226 | 116 | 36
  Week 48 | 57.1 | 26.7 | 25.0
  Week 60: number analyzed (Participants) | 211 | 110 | 35
  Week 60 | 60.2 | 30.0 | 42.9
  Week 72: number analyzed (Participants) | 204 | 103 | 33
  Week 72 | 56.4 | 29.1 | 36.4
  Week 84: number analyzed (Participants) | 204 | 95 | 33
  Week 84 | 60.3 | 29.5 | 54.5
  Week 96: number analyzed (Participants) | 199 | 94 | 33
  Week 96 | 57.3 | 34.0 | 42.4
  Week 108: number analyzed (Participants) | 192 | 91 | 34
  Week 108 | 59.9 | 31.9 | 47.1
  Week 120: number analyzed (Participants) | 187 | 88 | 29
  Week 120 | 59.4 | 30.7 | 62.1
  Week 132: number analyzed (Participants) | 178 | 80 | 29
  Week 132 | 61.8 | 33.8 | 48.3
  Week 144: number analyzed (Participants) | 172 | 73 | 28
  Week 144 | 57.6 | 34.2 | 39.3
  Week 156: number analyzed (Participants) | 173 | 72 | 27
  Week 156 | 64.7 | 38.9 | 55.6
  Week 168: number analyzed (Participants) | 170 | 71 | 29
  Week 168 | 62.9 | 42.3 | 58.6
  Week 180: number analyzed (Participants) | 176 | 71 | 29
  Week 180 | 59.1 | 29.6 | 48.3
  Week 192: number analyzed (Participants) | 163 | 69 | 27
  Week 192 | 62.0 | 31.9 | 48.1
  Week 204: number analyzed (Participants) | 163 | 68 | 29
  Week 204 | 65.0 | 42.6 | 58.6
  Week 216: number analyzed (Participants) | 159 | 62 | 28
  Week 216 | 59.1 | 41.9 | 46.4
  Week 228: number analyzed (Participants) | 150 | 56 | 28
  Week 228 | 60.0 | 39.3 | 60.7
  Week 240: number analyzed (Participants) | 151 | 62 | 28
  Week 240 | 66.2 | 38.7 | 46.4
  Week 252: number analyzed (Participants) | 143 | 58 | 28
  Week 252 | 62.9 | 29.3 | 50.0
  Week 264: number analyzed (Participants) | 135 | 54 | 28
  Week 264 | 58.5 | 37.0 | 57.1
  Week 276: number analyzed (Participants) | 127 | 52 | 25
  Week 276 | 66.1 | 34.6 | 48.0
  Week 288: number analyzed (Participants) | 132 | 52 | 27
  Week 288 | 65.9 | 44.2 | 44.4
  Week 300: number analyzed (Participants) | 125 | 51 | 23
  Week 300 | 60.8 | 41.2 | 43.5
  Week 312: number analyzed (Participants) | 130 | 48 | 27
  Week 312 | 63.1 | 39.6 | 55.6

4. Primary Outcome: Percentage of Participants With Satisfactory Humoral Response to PCV-13 Four Weeks After Vaccination
Description: Satisfactory humoral response is defined as greater than or equal to 2-fold increase in antibody concentration from the vaccination Baseline in at least 6 out of the 12 pneumococcal antigens 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F).
Time Frame: Vaccination Baseline (defined as the last non-missing observation on or before the date of receiving PCV-13 vaccination) and 4 weeks after vaccination
Population: The sub-study full analysis set (FAS) included all participants enrolled in the sub-study who received PCV-13 vaccination and at least 1 dose of upadacitinib 15 mg or 30 mg after vaccination during the sub-study. Analysis includes participants with available data at the Week 4 visit of the sub-study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Upadacitinib 15 mg + PCV-13: Participants receiving 15 mg upadacitinib QD were administered a single-dose of pneumococcal 13-valent conjugate vaccine (PCV-13).
- Upadacitinib 30 mg + PCV-13: Participants receiving 30 mg upadacitinib QD were administered a single-dose of pneumococcal 13-valent conjugate vaccine (PCV-13).
Arm/Group | Upadacitinib 15 mg + PCV-13 | Upadacitinib 30 mg + PCV-13
Number analyzed (Participants) | 83 | 23
percentage of participants | 67.5 [57.4 to 77.5] | 56.5 [36.3 to 76.8]

5. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on Disease Activity Score-28 (DAS28[CRP]) Over Time
Description: The DAS28(CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (measured on a VAS from 0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 (CRP) range from 0 to approximately 10, where higher scores indicate more disease activity.
  LDA is defined as a DAS28(CRP) score ≤ 3.2.
Time Frame: Weeks 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, and 312
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 279 | 146 | 37
  Week 6 | 70.3 | 43.2 | 43.2
  Week 12: number analyzed (Participants) | 272 | 145 | 37
  Week 12 | 77.9 | 43.4 | 43.2
  Week 24: number analyzed (Participants) | 255 | 134 | 36
  Week 24 | 82.4 | 48.5 | 52.8
  Week 36: number analyzed (Participants) | 246 | 128 | 36
  Week 36 | 80.5 | 50.8 | 55.6
  Week 48: number analyzed (Participants) | 228 | 118 | 37
  Week 48 | 86.8 | 54.2 | 56.8
  Week 60: number analyzed (Participants) | 218 | 110 | 36
  Week 60 | 86.2 | 56.4 | 66.7
  Week 72: number analyzed (Participants) | 203 | 104 | 33
  Week 72 | 84.7 | 51.0 | 69.7
  Week 84: number analyzed (Participants) | 207 | 98 | 34
  Week 84 | 88.9 | 60.2 | 85.3
  Week 96: number analyzed (Participants) | 205 | 97 | 34
  Week 96 | 82.4 | 64.9 | 79.4
  Week 108: number analyzed (Participants) | 195 | 92 | 34
  Week 108 | 88.2 | 66.3 | 70.6
  Week 120: number analyzed (Participants) | 185 | 87 | 31
  Week 120 | 85.9 | 69.0 | 77.4
  Week 132: number analyzed (Participants) | 167 | 77 | 31
  Week 132 | 88.6 | 70.1 | 87.1
  Week 144: number analyzed (Participants) | 169 | 70 | 28
  Week 144 | 85.2 | 68.6 | 82.1
  Week 156: number analyzed (Participants) | 166 | 67 | 29
  Week 156 | 86.1 | 74.6 | 86.2
  Week 168: number analyzed (Participants) | 160 | 69 | 30
  Week 168 | 90.0 | 78.3 | 80.0
  Week 180: number analyzed (Participants) | 178 | 69 | 30
  Week 180 | 90.4 | 69.6 | 80.0
  Week 192: number analyzed (Participants) | 169 | 72 | 27
  Week 192 | 89.3 | 75.0 | 96.3
  Week 204: number analyzed (Participants) | 166 | 70 | 30
  Week 204 | 88.6 | 61.4 | 83.3
  Week 216: number analyzed (Participants) | 159 | 64 | 28
  Week 216 | 89.9 | 70.3 | 82.1
  Week 228: number analyzed (Participants) | 151 | 55 | 29
  Week 228 | 89.4 | 70.9 | 86.2
  Week 240: number analyzed (Participants) | 153 | 62 | 29
  Week 240 | 89.5 | 75.8 | 86.2
  Week 252: number analyzed (Participants) | 145 | 58 | 31
  Week 252 | 91.7 | 67.2 | 83.9
  Week 264: number analyzed (Participants) | 130 | 53 | 28
  Week 264 | 86.2 | 67.9 | 82.1
  Week 276: number analyzed (Participants) | 121 | 54 | 25
  Week 276 | 91.7 | 74.1 | 72.0
  Week 288: number analyzed (Participants) | 106 | 46 | 25
  Week 288 | 90.6 | 71.7 | 76.0
  Week 300: number analyzed (Participants) | 101 | 37 | 20
  Week 300 | 94.1 | 67.6 | 80.0
  Week 312: number analyzed (Participants) | 116 | 48 | 27
  Week 312 | 84.5 | 68.8 | 70.4

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on Disease Activity Score-28 (DAS28[CRP]) Over Time
Description: The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (measured on a VAS from 0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 (CRP) range from 0 to approximately 10, where higher scores indicate more disease activity.
  Clinical remission is defined as a DAS28(CRP) score < 2.6.
Time Frame: as for outcome 5
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 279 | 146 | 37
  Week 6 | 53.0 | 21.2 | 29.7
  Week 12: number analyzed (Participants) | 272 | 145 | 37
  Week 12 | 56.6 | 25.5 | 27.0
  Week 24: number analyzed (Participants) | 255 | 134 | 36
  Week 24 | 60.8 | 31.3 | 38.9
  Week 36: number analyzed (Participants) | 246 | 128 | 36
  Week 36 | 65.0 | 35.2 | 50.0
  Week 48: number analyzed (Participants) | 228 | 118 | 37
  Week 48 | 66.2 | 36.4 | 35.1
  Week 60: number analyzed (Participants) | 218 | 110 | 36
  Week 60 | 72.9 | 38.2 | 50.0
  Week 72: number analyzed (Participants) | 203 | 104 | 33
  Week 72 | 69.0 | 35.6 | 51.5
  Week 84: number analyzed (Participants) | 207 | 98 | 34
  Week 84 | 72.0 | 36.7 | 52.9
  Week 96: number analyzed (Participants) | 205 | 97 | 34
  Week 96 | 71.7 | 45.4 | 52.9
  Week 108: number analyzed (Participants) | 195 | 92 | 34
  Week 108 | 74.4 | 42.4 | 47.1
  Week 120: number analyzed (Participants) | 185 | 87 | 31
  Week 120 | 74.1 | 49.4 | 45.2
  Week 132: number analyzed (Participants) | 167 | 77 | 31
  Week 132 | 73.7 | 40.3 | 61.3
  Week 144: number analyzed (Participants) | 169 | 70 | 28
  Week 144 | 71.0 | 44.3 | 60.7
  Week 156: number analyzed (Participants) | 166 | 67 | 29
  Week 156 | 74.7 | 50.7 | 65.5
  Week 168: number analyzed (Participants) | 160 | 69 | 30
  Week 168 | 77.5 | 49.3 | 66.7
  Week 180: number analyzed (Participants) | 178 | 69 | 30
  Week 180 | 75.3 | 44.9 | 56.7
  Week 192: number analyzed (Participants) | 169 | 72 | 27
  Week 192 | 76.9 | 47.2 | 55.6
  Week 204: number analyzed (Participants) | 166 | 70 | 30
  Week 204 | 77.1 | 47.1 | 76.7
  Week 216: number analyzed (Participants) | 159 | 64 | 28
  Week 216 | 79.2 | 56.3 | 53.6
  Week 228: number analyzed (Participants) | 151 | 55 | 29
  Week 228 | 80.8 | 49.1 | 69.0
  Week 240: number analyzed (Participants) | 153 | 62 | 29
  Week 240 | 75.2 | 50.0 | 69.0
  Week 252: number analyzed (Participants) | 145 | 58 | 31
  Week 252 | 80.7 | 44.8 | 58.1
  Week 264: number analyzed (Participants) | 130 | 53 | 28
  Week 264 | 73.8 | 39.6 | 67.9
  Week 276: number analyzed (Participants) | 121 | 54 | 25
  Week 276 | 76.9 | 50.0 | 52.0
  Week 288: number analyzed (Participants) | 106 | 46 | 25
  Week 288 | 74.5 | 47.8 | 48.0
  Week 300: number analyzed (Participants) | 101 | 37 | 20
  Week 300 | 75.2 | 43.2 | 55.0
  Week 312: number analyzed (Participants) | 116 | 48 | 27
  Week 312 | 72.4 | 45.8 | 63.0

7. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on Clinical Disease Activity Index (CDAI) Over Time
Description: The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm, and Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity.
  LDA is defined as a CDAI score ≤ 10.
Time Frame: as for outcome 5
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 274 | 142 | 37
  Week 6 | 65.3 | 35.2 | 35.1
  Week 12: number analyzed (Participants) | 273 | 141 | 34
  Week 12 | 71.1 | 39.7 | 32.4
  Week 24: number analyzed (Participants) | 254 | 133 | 35
  Week 24 | 80.3 | 46.6 | 51.4
  Week 36: number analyzed (Participants) | 243 | 126 | 35
  Week 36 | 77.8 | 44.4 | 57.1
  Week 48: number analyzed (Participants) | 230 | 118 | 36
  Week 48 | 83.0 | 50.8 | 38.9
  Week 60: number analyzed (Participants) | 218 | 107 | 36
  Week 60 | 85.8 | 58.9 | 63.9
  Week 72: number analyzed (Participants) | 200 | 104 | 33
  Week 72 | 85.5 | 46.2 | 60.6
  Week 84: number analyzed (Participants) | 205 | 97 | 32
  Week 84 | 84.4 | 52.6 | 75.0
  Week 96: number analyzed (Participants) | 198 | 96 | 33
  Week 96 | 81.3 | 63.5 | 57.6
  Week 108: number analyzed (Participants) | 194 | 86 | 33
  Week 108 | 85.1 | 67.4 | 54.5
  Week 120: number analyzed (Participants) | 188 | 88 | 31
  Week 120 | 87.2 | 67.0 | 77.4
  Week 132: number analyzed (Participants) | 182 | 80 | 30
  Week 132 | 87.4 | 72.5 | 76.7
  Week 144: number analyzed (Participants) | 181 | 75 | 28
  Week 144 | 88.4 | 68.0 | 78.6
  Week 156: number analyzed (Participants) | 178 | 71 | 28
  Week 156 | 88.8 | 73.2 | 71.4
  Week 168: number analyzed (Participants) | 173 | 73 | 30
  Week 168 | 90.8 | 82.2 | 83.3
  Week 180: number analyzed (Participants) | 179 | 69 | 30
  Week 180 | 88.3 | 73.9 | 76.7
  Week 192: number analyzed (Participants) | 168 | 70 | 29
  Week 192 | 88.1 | 70.0 | 79.3
  Week 204: number analyzed (Participants) | 164 | 70 | 29
  Week 204 | 89.0 | 71.4 | 82.8
  Week 216: number analyzed (Participants) | 158 | 64 | 28
  Week 216 | 88.6 | 70.3 | 78.6
  Week 228: number analyzed (Participants) | 149 | 56 | 29
  Week 228 | 89.3 | 67.9 | 79.3
  Week 240: number analyzed (Participants) | 153 | 62 | 29
  Week 240 | 87.6 | 72.6 | 75.9
  Week 252: number analyzed (Participants) | 146 | 57 | 31
  Week 252 | 89.0 | 73.7 | 74.2
  Week 264: number analyzed (Participants) | 133 | 54 | 29
  Week 264 | 83.5 | 63.0 | 75.9
  Week 276: number analyzed (Participants) | 129 | 53 | 28
  Week 276 | 87.6 | 67.9 | 67.9
  Week 288: number analyzed (Participants) | 134 | 51 | 28
  Week 288 | 90.3 | 74.5 | 75.0
  Week 300: number analyzed (Participants) | 127 | 50 | 24
  Week 300 | 89.8 | 72.0 | 70.8
  Week 312: number analyzed (Participants) | 127 | 47 | 26
  Week 312 | 86.6 | 70.2 | 73.1

8. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on Clinical Disease Activity Index (CDAI) Over Time
Description: The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm, and Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity.
  Clinical remission is defined as a CDAI score ≤ 2.8.
Time Frame: as for outcome 5
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 274 | 142 | 37
  Week 6 | 23.4 | 4.9 | 10.8
  Week 12: number analyzed (Participants) | 273 | 141 | 34
  Week 12 | 26.4 | 6.4 | 8.8
  Week 24: number analyzed (Participants) | 254 | 133 | 35
  Week 24 | 28.3 | 12.8 | 14.3
  Week 36: number analyzed (Participants) | 243 | 126 | 35
  Week 36 | 32.5 | 9.5 | 17.1
  Week 48: number analyzed (Participants) | 230 | 118 | 36
  Week 48 | 34.8 | 11.0 | 11.1
  Week 60: number analyzed (Participants) | 218 | 107 | 36
  Week 60 | 43.1 | 13.1 | 22.2
  Week 72: number analyzed (Participants) | 200 | 104 | 33
  Week 72 | 43.5 | 12.5 | 9.1
  Week 84: number analyzed (Participants) | 205 | 97 | 32
  Week 84 | 43.4 | 12.4 | 18.8
  Week 96: number analyzed (Participants) | 198 | 96 | 33
  Week 96 | 40.4 | 15.6 | 21.2
  Week 108: number analyzed (Participants) | 194 | 86 | 33
  Week 108 | 44.8 | 16.3 | 18.2
  Week 120: number analyzed (Participants) | 188 | 88 | 31
  Week 120 | 43.6 | 12.5 | 22.6
  Week 132: number analyzed (Participants) | 182 | 80 | 30
  Week 132 | 46.7 | 18.8 | 33.3
  Week 144: number analyzed (Participants) | 181 | 75 | 28
  Week 144 | 38.1 | 14.7 | 28.6
  Week 156: number analyzed (Participants) | 178 | 71 | 28
  Week 156 | 47.2 | 14.1 | 32.1
  Week 168: number analyzed (Participants) | 173 | 73 | 30
  Week 168 | 48.6 | 20.5 | 33.3
  Week 180: number analyzed (Participants) | 179 | 69 | 30
  Week 180 | 48.0 | 15.9 | 20.0
  Week 192: number analyzed (Participants) | 168 | 70 | 29
  Week 192 | 46.4 | 18.6 | 24.1
  Week 204: number analyzed (Participants) | 164 | 70 | 29
  Week 204 | 51.2 | 20.0 | 34.5
  Week 216: number analyzed (Participants) | 158 | 64 | 28
  Week 216 | 46.2 | 21.9 | 28.6
  Week 228: number analyzed (Participants) | 149 | 56 | 29
  Week 228 | 44.3 | 25.0 | 31.0
  Week 240: number analyzed (Participants) | 153 | 62 | 29
  Week 240 | 51.6 | 24.2 | 31.0
  Week 252: number analyzed (Participants) | 146 | 57 | 31
  Week 252 | 52.7 | 19.3 | 22.6
  Week 264: number analyzed (Participants) | 133 | 54 | 29
  Week 264 | 48.1 | 20.4 | 17.2
  Week 276: number analyzed (Participants) | 129 | 53 | 28
  Week 276 | 53.5 | 24.5 | 28.6
  Week 288: number analyzed (Participants) | 134 | 51 | 28
  Week 288 | 51.5 | 25.5 | 28.6
  Week 300: number analyzed (Participants) | 127 | 50 | 24
  Week 300 | 51.2 | 22.0 | 29.2
  Week 312: number analyzed (Participants) | 127 | 47 | 26
  Week 312 | 50.4 | 27.7 | 34.6

9. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on Simplified Disease Activity Index (SDAI) Over Time
Description: The simplified disease activity index (SDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm, Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm and hsCRP (mg/dL). The total SDAI score ranges from 0 to 86 with higher scores indicating higher disease activity.
  LDA is defined as a SDAI score ≤ 11.0.
Time Frame: as for outcome 5
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 273 | 142 | 37
  Week 6 | 54.2 | 25.4 | 32.4
  Week 12: number analyzed (Participants) | 270 | 141 | 34
  Week 12 | 61.1 | 33.3 | 23.5
  Week 24: number analyzed (Participants) | 253 | 133 | 35
  Week 24 | 66.8 | 33.1 | 48.6
  Week 36: number analyzed (Participants) | 242 | 126 | 35
  Week 36 | 67.8 | 34.9 | 48.6
  Week 48: number analyzed (Participants) | 228 | 118 | 36
  Week 48 | 73.7 | 38.1 | 41.7
  Week 60: number analyzed (Participants) | 218 | 107 | 36
  Week 60 | 72.9 | 41.1 | 61.1
  Week 72: number analyzed (Participants) | 200 | 104 | 33
  Week 72 | 71.5 | 36.5 | 51.5
  Week 84: number analyzed (Participants) | 205 | 97 | 32
  Week 84 | 74.6 | 40.2 | 62.5
  Week 96: number analyzed (Participants) | 198 | 96 | 33
  Week 96 | 71.2 | 45.8 | 51.5
  Week 108: number analyzed (Participants) | 194 | 86 | 33
  Week 108 | 75.8 | 51.2 | 54.5
  Week 120: number analyzed (Participants) | 185 | 87 | 31
  Week 120 | 74.6 | 55.2 | 64.5
  Week 132: number analyzed (Participants) | 166 | 76 | 30
  Week 132 | 77.7 | 43.4 | 66.7
  Week 144: number analyzed (Participants) | 167 | 70 | 28
  Week 144 | 70.7 | 44.3 | 67.9
  Week 156: number analyzed (Participants) | 164 | 65 | 28
  Week 156 | 75.0 | 58.5 | 64.3
  Week 168: number analyzed (Participants) | 157 | 69 | 30
  Week 168 | 75.8 | 59.4 | 66.7
  Week 180: number analyzed (Participants) | 178 | 68 | 30
  Week 180 | 78.7 | 55.9 | 53.3
  Week 192: number analyzed (Participants) | 168 | 70 | 27
  Week 192 | 76.2 | 52.9 | 66.7
  Week 204: number analyzed (Participants) | 164 | 70 | 29
  Week 204 | 71.3 | 52.9 | 79.3
  Week 216: number analyzed (Participants) | 157 | 64 | 28
  Week 216 | 79.0 | 56.3 | 57.1
  Week 228: number analyzed (Participants) | 149 | 55 | 29
  Week 228 | 77.2 | 56.4 | 69.0
  Week 240: number analyzed (Participants) | 153 | 62 | 29
  Week 240 | 74.5 | 50.0 | 69.0
  Week 252: number analyzed (Participants) | 143 | 57 | 31
  Week 252 | 79.0 | 52.6 | 61.3
  Week 264: number analyzed (Participants) | 128 | 52 | 28
  Week 264 | 71.1 | 51.9 | 67.9
  Week 276: number analyzed (Participants) | 121 | 53 | 25
  Week 276 | 78.5 | 56.6 | 56.0
  Week 288: number analyzed (Participants) | 106 | 46 | 25
  Week 288 | 74.5 | 56.5 | 68.0
  Week 300: number analyzed (Participants) | 101 | 36 | 19
  Week 300 | 78.2 | 50.0 | 63.2
  Week 312: number analyzed (Participants) | 111 | 45 | 26
  Week 312 | 72.1 | 48.9 | 65.4

10. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on Simplified Disease Activity Index (SDAI) Over Time
Description: The simplified disease activity index (SDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm, Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm and hsCRP (mg/dL). The total SDAI score ranges from 0 to 86 with higher scores indicating higher disease activity.
  Clinical remission is defined as a SDAI score ≤ 3.3.
Time Frame: as for outcome 5
Population: Open-label treated population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
percentage of participants
  Week 6: number analyzed (Participants) | 273 | 142 | 37
  Week 6 | 15.0 | 4.2 | 2.7
  Week 12: number analyzed (Participants) | 270 | 141 | 34
  Week 12 | 17.8 | 2.8 | 5.9
  Week 24: number analyzed (Participants) | 253 | 133 | 35
  Week 24 | 18.2 | 6.0 | 11.4
  Week 36: number analyzed (Participants) | 242 | 126 | 35
  Week 36 | 23.6 | 4.0 | 8.6
  Week 48: number analyzed (Participants) | 228 | 118 | 36
  Week 48 | 25.9 | 7.6 | 8.3
  Week 60: number analyzed (Participants) | 218 | 107 | 36
  Week 60 | 32.6 | 12.1 | 13.9
  Week 72: number analyzed (Participants) | 200 | 104 | 33
  Week 72 | 31.0 | 9.6 | 9.1
  Week 84: number analyzed (Participants) | 205 | 97 | 32
  Week 84 | 32.2 | 8.2 | 12.5
  Week 96: number analyzed (Participants) | 198 | 96 | 33
  Week 96 | 28.8 | 13.5 | 18.2
  Week 108: number analyzed (Participants) | 194 | 86 | 33
  Week 108 | 31.4 | 10.5 | 12.1
  Week 120: number analyzed (Participants) | 185 | 87 | 31
  Week 120 | 33.5 | 8.0 | 12.9
  Week 132: number analyzed (Participants) | 166 | 76 | 30
  Week 132 | 33.1 | 10.5 | 20.0
  Week 144: number analyzed (Participants) | 167 | 70 | 28
  Week 144 | 26.3 | 5.7 | 14.3
  Week 156: number analyzed (Participants) | 164 | 65 | 28
  Week 156 | 33.5 | 7.7 | 28.6
  Week 168: number analyzed (Participants) | 157 | 69 | 30
  Week 168 | 31.8 | 11.6 | 26.7
  Week 180: number analyzed (Participants) | 178 | 68 | 30
  Week 180 | 33.1 | 10.3 | 13.3
  Week 192: number analyzed (Participants) | 168 | 70 | 27
  Week 192 | 32.7 | 12.9 | 14.8
  Week 204: number analyzed (Participants) | 164 | 70 | 29
  Week 204 | 37.2 | 11.4 | 24.1
  Week 216: number analyzed (Participants) | 157 | 64 | 28
  Week 216 | 32.5 | 10.9 | 10.7
  Week 228: number analyzed (Participants) | 149 | 55 | 29
  Week 228 | 30.9 | 16.4 | 24.1
  Week 240: number analyzed (Participants) | 153 | 62 | 29
  Week 240 | 34.0 | 14.5 | 10.3
  Week 252: number analyzed (Participants) | 143 | 57 | 31
  Week 252 | 39.9 | 12.3 | 16.1
  Week 264: number analyzed (Participants) | 128 | 52 | 28
  Week 264 | 32.8 | 11.5 | 7.1
  Week 276: number analyzed (Participants) | 121 | 53 | 25
  Week 276 | 35.5 | 17.0 | 20.0
  Week 288: number analyzed (Participants) | 106 | 46 | 25
  Week 288 | 35.8 | 19.6 | 8.0
  Week 300: number analyzed (Participants) | 101 | 36 | 19
  Week 300 | 34.7 | 16.7 | 26.3
  Week 312: number analyzed (Participants) | 111 | 45 | 26
  Week 312 | 30.6 | 15.6 | 26.9

11. Secondary Outcome: Change From Baseline in Disease Activity Score Based on CRP (DAS28 [CRP]) Over Time
Description: The disease activity score-28-CRP (DAS28 [CRP]) assesses RA disease activity based on a continuous scale of combined measures of 28 tender joint counts (TJC28), 28 swollen joint counts (SJC28), C-reactive protein (CRP), and the patient global assessment of disease activity (measured on a visual analog scale from 0 to 100 mm). DAS28(CRP) scores range from 0 to approximately 10 where higher scores indicate more disease activity. A negative change from Baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: as for outcome 1
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 305 | 146 | 37
score on a scale
  Week 6: number analyzed (Participants) | 278 | 144 | 36
  Week 6 | -2.9 (1.21) | -2.4 (1.28) | -2.5 (1.01)
  Week 12: number analyzed (Participants) | 271 | 143 | 36
  Week 12 | -3.1 (1.14) | -2.5 (1.27) | -2.5 (1.03)
  Week 24: number analyzed (Participants) | 254 | 132 | 35
  Week 24 | -3.2 (1.07) | -2.7 (1.36) | -2.7 (1.22)
  Week 36: number analyzed (Participants) | 245 | 126 | 35
  Week 36 | -3.2 (1.20) | -2.9 (1.11) | -3.0 (1.17)
  Week 48: number analyzed (Participants) | 227 | 116 | 36
  Week 48 | -3.4 (1.20) | -2.9 (1.20) | -2.8 (0.97)
  Week 60: number analyzed (Participants) | 217 | 108 | 35
  Week 60 | -3.5 (1.15) | -2.9 (1.07) | -3.1 (0.98)
  Week 72: number analyzed (Participants) | 202 | 102 | 32
  Week 72 | -3.5 (1.03) | -2.9 (1.24) | -3.1 (0.88)
  Week 84: number analyzed (Participants) | 206 | 96 | 33
  Week 84 | -3.5 (1.06) | -2.9 (1.28) | -3.3 (0.62)
  Week 96: number analyzed (Participants) | 204 | 95 | 33
  Week 96 | -3.4 (1.11) | -3.1 (1.21) | -3.2 (0.98)
  Week 108: number analyzed (Participants) | 195 | 91 | 33
  Week 108 | -3.5 (1.09) | -3.1 (1.24) | -3.1 (0.94)
  Week 120: number analyzed (Participants) | 185 | 86 | 30
  Week 120 | -3.5 (1.08) | -3.1 (1.29) | -3.2 (0.86)
  Week 132: number analyzed (Participants) | 167 | 77 | 30
  Week 132 | -3.5 (1.02) | -3.1 (1.23) | -3.3 (1.02)
  Week 144: number analyzed (Participants) | 169 | 70 | 27
  Week 144 | -3.4 (1.13) | -3.0 (1.18) | -3.4 (1.04)
  Week 156: number analyzed (Participants) | 166 | 67 | 28
  Week 156 | -3.5 (1.13) | -3.1 (1.11) | -3.6 (1.00)
  Week 168: number analyzed (Participants) | 160 | 68 | 29
  Week 168 | -3.6 (1.17) | -3.2 (1.23) | -3.6 (1.08)
  Week 180: number analyzed (Participants) | 178 | 68 | 29
  Week 180 | -3.6 (1.10) | -3.2 (1.24) | -3.5 (1.13)
  Week 192: number analyzed (Participants) | 169 | 72 | 26
  Week 192 | -3.6 (1.15) | -3.2 (1.31) | -3.6 (1.06)
  Week 204: number analyzed (Participants) | 166 | 70 | 29
  Week 204 | -3.6 (1.13) | -3.1 (1.32) | -3.7 (1.13)
  Week 216: number analyzed (Participants) | 159 | 64 | 27
  Week 216 | -3.6 (1.13) | -3.2 (1.15) | -3.5 (1.02)
  Week 228: number analyzed (Participants) | 151 | 54 | 28
  Week 228 | -3.6 (1.12) | -3.3 (1.37) | -3.7 (0.91)
  Week 240: number analyzed (Participants) | 153 | 61 | 28
  Week 240 | -3.7 (1.12) | -3.2 (1.30) | -3.5 (0.91)
  Week 252: number analyzed (Participants) | 145 | 58 | 30
  Week 252 | -3.7 (1.20) | -3.3 (1.18) | -3.3 (1.04)
  Week 264: number analyzed (Participants) | 130 | 53 | 27
  Week 264 | -3.5 (1.25) | -3.1 (1.24) | -3.4 (1.01)
  Week 276: number analyzed (Participants) | 121 | 53 | 24
  Week 276 | -3.7 (1.01) | -3.1 (1.22) | -3.5 (0.90)
  Week 288: number analyzed (Participants) | 106 | 45 | 24
  Week 288 | -3.7 (1.08) | -3.3 (1.44) | -3.2 (0.75)
  Week 300: number analyzed (Participants) | 101 | 36 | 19
  Week 300 | -3.7 (1.00) | -3.0 (1.38) | -3.4 (0.81)
  Week 312: number analyzed (Participants) | 116 | 47 | 26
  Week 312 | -3.5 (1.10) | -3.2 (1.25) | -3.2 (1.04)

12. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Over Time
Description: The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm, and Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. A negative change from Baseline indicates improvement in disease activity.
Time Frame: as for outcome 1
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 297 | 144 | 37
score on a scale
  Week 6: number analyzed (Participants) | 265 | 138 | 36
  Week 6 | -30.0 (12.49) | -27.5 (13.54) | -27.2 (11.42)
  Week 12: number analyzed (Participants) | 265 | 137 | 33
  Week 12 | -31.6 (11.82) | -28.4 (13.87) | -27.9 (11.12)
  Week 24: number analyzed (Participants) | 246 | 129 | 34
  Week 24 | -32.6 (11.81) | -30.6 (13.59) | -29.6 (11.45)
  Week 36: number analyzed (Participants) | 236 | 122 | 34
  Week 36 | -32.2 (12.43) | -31.4 (12.67) | -29.6 (11.63)
  Week 48: number analyzed (Participants) | 222 | 114 | 35
  Week 48 | -34.0 (12.84) | -31.8 (13.35) | -29.1 (10.82)
  Week 60: number analyzed (Participants) | 210 | 103 | 35
  Week 60 | -34.7 (12.52) | -32.4 (12.18) | -32.2 (12.09)
  Week 72: number analyzed (Participants) | 192 | 100 | 32
  Week 72 | -34.3 (11.71) | -32.3 (13.33) | -31.8 (10.88)
  Week 84: number analyzed (Participants) | 197 | 93 | 31
  Week 84 | -34.9 (12.08) | -31.0 (13.36) | -33.5 (9.66)
  Week 96: number analyzed (Participants) | 191 | 92 | 32
  Week 96 | -33.4 (11.71) | -32.1 (12.37) | -31.3 (10.86)
  Week 108: number analyzed (Participants) | 187 | 83 | 32
  Week 108 | -34.5 (11.83) | -32.4 (12.79) | -32.3 (10.81)
  Week 120: number analyzed (Participants) | 181 | 85 | 30
  Week 120 | -34.8 (11.87) | -32.3 (12.94) | -34.0 (10.75)
  Week 132: number analyzed (Participants) | 175 | 79 | 29
  Week 132 | -35.0 (12.24) | -32.7 (12.39) | -34.5 (12.14)
  Week 144: number analyzed (Participants) | 174 | 74 | 27
  Week 144 | -35.0 (12.21) | -33.1 (12.67) | -36.2 (12.03)
  Week 156: number analyzed (Participants) | 171 | 69 | 27
  Week 156 | -35.6 (12.24) | -33.6 (12.25) | -36.1 (11.80)
  Week 168: number analyzed (Participants) | 166 | 70 | 29
  Week 168 | -36.2 (13.01) | -33.8 (12.97) | -37.6 (13.08)
  Week 180: number analyzed (Participants) | 172 | 66 | 29
  Week 180 | -35.5 (12.60) | -34.0 (12.13) | -36.9 (12.07)
  Week 192: number analyzed (Participants) | 161 | 68 | 28
  Week 192 | -35.6 (12.25) | -34.0 (12.89) | -38.6 (11.76)
  Week 204: number analyzed (Participants) | 157 | 68 | 28
  Week 204 | -36.0 (12.36) | -33.8 (13.69) | -37.9 (12.59)
  Week 216: number analyzed (Participants) | 151 | 62 | 27
  Week 216 | -35.8 (13.19) | -33.9 (11.87) | -37.3 (11.62)
  Week 228: number analyzed (Participants) | 143 | 53 | 28
  Week 228 | -35.6 (12.68) | -35.5 (13.31) | -37.9 (11.55)
  Week 240: number analyzed (Participants) | 146 | 59 | 28
  Week 240 | -36.4 (12.95) | -34.7 (13.02) | -35.8 (11.07)
  Week 252: number analyzed (Participants) | 139 | 55 | 30
  Week 252 | -35.9 (13.41) | -35.3 (12.58) | -34.3 (11.71)
  Week 264: number analyzed (Participants) | 126 | 52 | 28
  Week 264 | -35.5 (13.66) | -33.2 (12.38) | -33.5 (12.49)
  Week 276: number analyzed (Participants) | 122 | 50 | 27
  Week 276 | -36.5 (12.59) | -33.6 (12.16) | -34.7 (11.92)
  Week 288: number analyzed (Participants) | 129 | 48 | 27
  Week 288 | -36.9 (13.22) | -35.3 (14.34) | -33.5 (10.25)
  Week 300: number analyzed (Participants) | 120 | 47 | 23
  Week 300 | -36.0 (12.17) | -32.9 (11.86) | -34.6 (11.27)
  Week 312: number analyzed (Participants) | 120 | 44 | 25
  Week 312 | -35.9 (12.43) | -34.4 (12.63) | -34.0 (11.62)

13. Secondary Outcome: Change From Baseline in SimplifiedDisease Activity Index (SDAI) Over Time
Description: The simplified disease activity index (SDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm, Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10 cm and hsCRP (mg/dL). The total SDAI score ranges from 0 to 86 with higher scores indicating higher disease activity. A negative change from Baseline indicates improvement in disease activity.
Time Frame: as for outcome 1
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 297 | 144 | 37
score on a scale
  Week 6: number analyzed (Participants) | 264 | 138 | 36
  Week 6 | -38.8 (25.57) | -37.2 (27.36) | -40.8 (29.76)
  Week 12: number analyzed (Participants) | 262 | 137 | 33
  Week 12 | -40.6 (24.84) | -38.6 (26.09) | -41.7 (30.24)
  Week 24: number analyzed (Participants) | 245 | 129 | 34
  Week 24 | -42.0 (23.35) | -36.7 (43.09) | -38.2 (33.62)
  Week 36: number analyzed (Participants) | 235 | 122 | 34
  Week 36 | -41.8 (25.10) | -41.6 (25.59) | -44.5 (31.98)
  Week 48: number analyzed (Participants) | 220 | 114 | 35
  Week 48 | -42.9 (23.24) | -41.6 (25.26) | -44.6 (29.09)
  Week 60: number analyzed (Participants) | 210 | 103 | 35
  Week 60 | -44.3 (24.21) | -42.5 (24.51) | -41.4 (22.38)
  Week 72: number analyzed (Participants) | 192 | 100 | 32
  Week 72 | -43.4 (24.62) | -41.9 (27.31) | -41.8 (21.19)
  Week 84: number analyzed (Participants) | 197 | 93 | 31
  Week 84 | -42.7 (28.14) | -39.0 (31.94) | -44.7 (20.79)
  Week 96: number analyzed (Participants) | 191 | 92 | 32
  Week 96 | -42.0 (18.50) | -42.4 (27.17) | -43.2 (22.39)
  Week 108: number analyzed (Participants) | 187 | 83 | 32
  Week 108 | -43.6 (27.35) | -42.9 (24.31) | -44.0 (21.38)
  Week 120: number analyzed (Participants) | 178 | 84 | 30
  Week 120 | -42.7 (22.25) | -43.7 (25.88) | -43.4 (23.39)
  Week 132: number analyzed (Participants) | 165 | 76 | 29
  Week 132 | -43.4 (19.92) | -41.4 (27.64) | -44.2 (23.86)
  Week 144: number analyzed (Participants) | 166 | 70 | 27
  Week 144 | -41.7 (22.60) | -43.0 (29.91) | -46.0 (25.20)
  Week 156: number analyzed (Participants) | 163 | 64 | 27
  Week 156 | -42.8 (21.64) | -43.6 (29.88) | -48.0 (23.98)
  Week 168: number analyzed (Participants) | 156 | 67 | 29
  Week 168 | -43.7 (23.75) | -43.2 (28.55) | -46.4 (23.28)
  Week 180: number analyzed (Participants) | 171 | 65 | 29
  Week 180 | -45.6 (26.65) | -45.0 (27.57) | -47.2 (24.08)
  Week 192: number analyzed (Participants) | 161 | 68 | 26
  Week 192 | -44.7 (30.13) | -44.4 (27.94) | -48.5 (25.36)
  Week 204: number analyzed (Participants) | 157 | 68 | 28
  Week 204 | -44.1 (35.23) | -43.5 (28.81) | -47.6 (24.55)
  Week 216: number analyzed (Participants) | 150 | 62 | 27
  Week 216 | -47.3 (27.43) | -44.2 (26.69) | -47.4 (23.26)
  Week 228: number analyzed (Participants) | 143 | 52 | 28
  Week 228 | -46.0 (27.33) | -47.9 (28.86) | -48.6 (21.47)
  Week 240: number analyzed (Participants) | 146 | 59 | 28
  Week 240 | -46.8 (31.40) | -44.2 (29.63) | -45.0 (21.97)
  Week 252: number analyzed (Participants) | 136 | 55 | 30
  Week 252 | -45.9 (25.86) | -45.7 (29.98) | -44.3 (23.50)
  Week 264: number analyzed (Participants) | 121 | 50 | 27
  Week 264 | -44.9 (24.26) | -43.5 (30.06) | -44.4 (21.96)
  Week 276: number analyzed (Participants) | 114 | 50 | 24
  Week 276 | -46.3 (20.01) | -44.2 (26.93) | -47.4 (20.53)
  Week 288: number analyzed (Participants) | 105 | 44 | 24
  Week 288 | -47.1 (22.36) | -48.3 (30.14) | -41.6 (17.15)
  Week 300: number analyzed (Participants) | 98 | 34 | 18
  Week 300 | -47.4 (20.47) | -41.6 (26.38) | -42.7 (19.05)
  Week 312: number analyzed (Participants) | 110 | 43 | 25
  Week 312 | -45.8 (28.64) | -45.8 (28.89) | -41.2 (17.55)

14. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC68) Over Time
Description: Sixty-eight joints were assessed by an evaluator for tenderness or pain. The presence of tenderness was scored as a "1" and absence of tenderness as a "0". The total tender joint count is the sum of the scores, and ranges from 0 to 68 (worst).
Time Frame: as for outcome 1
Population: Open-label treated population with available data at each time point
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
joints
  Week 6: number analyzed (Participants) | 284 | 146 | 37
  Week 6 | -20.6 (12.81) | -21.3 (14.53) | -22.1 (12.90)
  Week 12: number analyzed (Participants) | 280 | 145 | 37
  Week 12 | -21.3 (12.47) | -22.5 (14.65) | -20.5 (11.18)
  Week 24: number analyzed (Participants) | 258 | 137 | 36
  Week 24 | -22.0 (12.96) | -23.9 (14.60) | -22.9 (12.17)
  Week 36: number analyzed (Participants) | 248 | 133 | 36
  Week 36 | -21.7 (12.58) | -24.2 (14.45) | -23.4 (13.56)
  Week 48: number analyzed (Participants) | 234 | 121 | 37
  Week 48 | -23.1 (13.61) | -24.1 (14.43) | -24.0 (13.13)
  Week 60: number analyzed (Participants) | 218 | 110 | 36
  Week 60 | -23.6 (13.56) | -25.0 (14.42) | -25.6 (13.54)
  Week 72: number analyzed (Participants) | 204 | 104 | 33
  Week 72 | -23.3 (13.06) | -24.3 (14.48) | -26.1 (13.12)
  Week 84: number analyzed (Participants) | 209 | 98 | 34
  Week 84 | -23.2 (12.71) | -23.4 (14.23) | -27.4 (13.32)
  Week 96: number analyzed (Participants) | 206 | 97 | 34
  Week 96 | -23.1 (12.90) | -23.9 (14.58) | -24.6 (11.94)
  Week 108: number analyzed (Participants) | 195 | 92 | 34
  Week 108 | -23.3 (12.62) | -23.7 (14.22) | -25.2 (12.31)
  Week 120: number analyzed (Participants) | 189 | 92 | 34
  Week 120 | -23.1 (13.13) | -23.9 (14.17) | -26.9 (12.72)
  Week 132: number analyzed (Participants) | 184 | 82 | 31
  Week 132 | -23.1 (12.79) | -23.7 (13.95) | -26.8 (13.74)
  Week 144: number analyzed (Participants) | 183 | 75 | 28
  Week 144 | -23.5 (13.28) | -23.8 (13.50) | -29.3 (13.19)
  Week 156: number analyzed (Participants) | 181 | 73 | 30
  Week 156 | -23.7 (13.21) | -23.9 (13.00) | -28.1 (13.63)
  Week 168: number analyzed (Participants) | 177 | 74 | 30
  Week 168 | -24.1 (13.82) | -24.4 (13.86) | -31.0 (14.12)
  Week 180: number analyzed (Participants) | 180 | 70 | 30
  Week 180 | -23.7 (13.60) | -24.9 (14.12) | -29.5 (12.96)
  Week 192: number analyzed (Participants) | 169 | 72 | 29
  Week 192 | -24.0 (13.75) | -24.4 (14.15) | -31.3 (13.80)
  Week 204: number analyzed (Participants) | 167 | 70 | 30
  Week 204 | -24.2 (13.77) | -23.6 (14.35) | -30.4 (14.53)
  Week 216: number analyzed (Participants) | 160 | 64 | 28
  Week 216 | -24.2 (13.82) | -24.1 (13.87) | -31.6 (13.80)
  Week 228: number analyzed (Participants) | 154 | 56 | 30
  Week 228 | -23.9 (13.57) | -26.6 (14.65) | -30.5 (13.69)
  Week 240: number analyzed (Participants) | 154 | 62 | 29
  Week 240 | -24.7 (14.09) | -25.6 (14.47) | -29.4 (14.28)
  Week 252: number analyzed (Participants) | 148 | 58 | 31
  Week 252 | -24.2 (13.78) | -25.6 (14.14) | -27.5 (13.26)
  Week 264: number analyzed (Participants) | 135 | 55 | 29
  Week 264 | -23.7 (13.56) | -23.7 (13.28) | -27.0 (13.76)
  Week 276: number analyzed (Participants) | 129 | 54 | 28
  Week 276 | -23.6 (13.55) | -23.9 (13.76) | -28.0 (14.41)
  Week 288: number analyzed (Participants) | 137 | 51 | 28
  Week 288 | -24.9 (14.42) | -25.7 (14.87) | -26.6 (14.42)
  Week 300: number analyzed (Participants) | 127 | 51 | 26
  Week 300 | -24.3 (14.04) | -24.5 (15.18) | -28.2 (14.10)
  Week 312: number analyzed (Participants) | 133 | 50 | 27
  Week 312 | -24.1 (13.82) | -23.2 (14.08) | -26.8 (14.48)

15. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC66) Over Time
Description: Sixty-six joints were assessed by an evaluator for swelling. The presence of swelling was scored as a "1" and absence of swelling as a "0". The total swollen joint count is the sum of the scores, and ranges from 0 to 66 (worst).
Time Frame: as for outcome 1
Population: Open-label treated population with available data at each time point
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
joints
  Week 6: number analyzed (Participants) | 284 | 146 | 37
  Week 6 | -12.8 (7.76) | -13.5 (10.89) | -14.5 (8.70)
  Week 12: number analyzed (Participants) | 280 | 145 | 37
  Week 12 | -13.7 (7.95) | -13.9 (11.26) | -13.5 (6.72)
  Week 24: number analyzed (Participants) | 258 | 137 | 36
  Week 24 | -14.2 (8.31) | -14.7 (10.87) | -15.7 (5.67)
  Week 36: number analyzed (Participants) | 248 | 133 | 36
  Week 36 | -14.1 (8.26) | -15.1 (10.39) | -15.6 (5.94)
  Week 48: number analyzed (Participants) | 234 | 121 | 37
  Week 48 | -15.3 (9.47) | -15.4 (11.19) | -16.0 (6.10)
  Week 60: number analyzed (Participants) | 218 | 110 | 36
  Week 60 | -15.6 (9.52) | -15.9 (11.83) | -17.4 (9.36)
  Week 72: number analyzed (Participants) | 204 | 104 | 33
  Week 72 | -15.1 (8.50) | -15.5 (10.47) | -17.0 (6.31)
  Week 84: number analyzed (Participants) | 209 | 98 | 34
  Week 84 | -15.6 (9.18) | -14.7 (9.96) | -17.0 (6.68)
  Week 96: number analyzed (Participants) | 206 | 97 | 34
  Week 96 | -15.3 (9.27) | -14.7 (9.48) | -16.6 (6.79)
  Week 108: number analyzed (Participants) | 195 | 92 | 34
  Week 108 | -15.2 (8.72) | -15.2 (10.17) | -16.6 (6.96)
  Week 120: number analyzed (Participants) | 189 | 89 | 31
  Week 120 | -15.6 (8.77) | -14.8 (9.06) | -17.5 (7.15)
  Week 132: number analyzed (Participants) | 184 | 82 | 31
  Week 132 | -15.7 (9.23) | -14.6 (9.79) | -17.3 (7.11)
  Week 144: number analyzed (Participants) | 183 | 75 | 28
  Week 144 | -15.9 (9.03) | -15.3 (9.81) | -18.6 (7.17)
  Week 156: number analyzed (Participants) | 181 | 73 | 30
  Week 156 | -16.1 (9.74) | -15.5 (9.53) | -17.5 (7.89)
  Week 168: number analyzed (Participants) | 177 | 74 | 30
  Week 168 | -16.9 (11.11) | -15.8 (10.51) | -20.0 (9.94)
  Week 180: number analyzed (Participants) | 180 | 70 | 30
  Week 180 | -16.6 (10.67) | -16.2 (10.61) | -20.0 (9.91)
  Week 192: number analyzed (Participants) | 169 | 72 | 29
  Week 192 | -16.4 (9.87) | -15.8 (9.23) | -20.7 (10.08)
  Week 204: number analyzed (Participants) | 167 | 70 | 30
  Week 204 | -16.7 (10.60) | -15.9 (9.53) | -19.6 (10.22)
  Week 216: number analyzed (Participants) | 160 | 64 | 28
  Week 216 | -16.6 (10.29) | -16.1 (8.86) | -20.4 (10.12)
  Week 228: number analyzed (Participants) | 154 | 56 | 30
  Week 228 | -16.2 (9.51) | -17.3 (10.79) | -19.8 (10.16)
  Week 240: number analyzed (Participants) | 154 | 62 | 29
  Week 240 | -16.8 (10.41) | -17.0 (10.43) | -18.8 (7.86)
  Week 252: number analyzed (Participants) | 148 | 58 | 31
  Week 252 | -16.8 (10.63) | -16.9 (9.37) | -18.1 (7.78)
  Week 264: number analyzed (Participants) | 135 | 55 | 29
  Week 264 | -17.7 (11.38) | -16.1 (8.72) | -18.3 (7.55)
  Week 276: number analyzed (Participants) | 129 | 54 | 28
  Week 276 | -17.8 (11.35) | -17.0 (10.60) | -18.9 (7.74)
  Week 288: number analyzed (Participants) | 137 | 51 | 28
  Week 288 | -17.4 (11.28) | -17.8 (11.76) | -18.7 (7.67)
  Week 300: number analyzed (Participants) | 127 | 51 | 26
  Week 300 | -16.7 (10.21) | -17.1 (10.31) | -19.3 (7.72)
  Week 312: number analyzed (Participants) | 133 | 50 | 27
  Week 312 | -16.7 (9.71) | -17.4 (10.41) | -18.6 (7.51)

16. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity Over Time
Description: The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a visual analog scale (VAS) from 0 to 100 mm, where 0 mm indicates no disease activity and 100 mm indicates severe disease activity
Time Frame: as for outcome 1
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 298 | 147 | 38
score on a scale
  Week 6: number analyzed (Participants) | 268 | 140 | 37
  Week 6 | -46.8 (20.58) | -35.5 (21.53) | -38.4 (24.08)
  Week 12: number analyzed (Participants) | 269 | 140 | 34
  Week 12 | -48.9 (20.45) | -39.1 (22.99) | -37.5 (21.78)
  Week 24: number analyzed (Participants) | 248 | 133 | 36
  Week 24 | -51.2 (18.71) | -42.5 (21.24) | -40.9 (22.79)
  Week 36: number analyzed (Participants) | 236 | 124 | 35
  Week 36 | -51.6 (19.08) | -42.7 (20.96) | -39.5 (24.20)
  Week 48: number analyzed (Participants) | 223 | 116 | 36
  Week 48 | -52.8 (19.12) | -45.6 (19.29) | -40.6 (20.97)
  Week 60: number analyzed (Participants) | 211 | 106 | 36
  Week 60 | -54.2 (16.44) | -47.1 (19.64) | -44.7 (24.33)
  Week 72: number analyzed (Participants) | 198 | 103 | 34
  Week 72 | -53.4 (17.46) | -45.9 (18.58) | -47.2 (18.47)
  Week 84: number analyzed (Participants) | 199 | 96 | 32
  Week 84 | -54.3 (16.44) | -43.4 (21.41) | -48.5 (17.25)
  Week 96: number analyzed (Participants) | 192 | 95 | 33
  Week 96 | -52.3 (17.69) | -45.7 (20.42) | -46.8 (20.97)
  Week 108: number analyzed (Participants) | 187 | 86 | 33
  Week 108 | -55.5 (16.72) | -45.9 (18.75) | -47.4 (21.09)
  Week 120: number analyzed (Participants) | 182 | 86 | 31
  Week 120 | -55.9 (16.38) | -48.6 (18.23) | -50.1 (21.51)
  Week 132: number analyzed (Participants) | 177 | 79 | 30
  Week 132 | -56.1 (16.60) | -50.1 (17.19) | -52.5 (20.62)
  Week 144: number analyzed (Participants) | 174 | 74 | 29
  Week 144 | -56.7 (15.79) | -48.2 (18.28) | -51.4 (19.66)
  Week 156: number analyzed (Participants) | 172 | 70 | 29
  Week 156 | -57.0 (16.90) | -48.9 (18.89) | -52.4 (19.49)
  Week 168: number analyzed (Participants) | 168 | 73 | 30
  Week 168 | -57.0 (15.94) | -51.9 (20.24) | -55.6 (21.25)
  Week 180: number analyzed (Participants) | 174 | 68 | 30
  Week 180 | -57.2 (17.11) | -53.0 (18.04) | -53.1 (19.34)
  Week 192: number analyzed (Participants) | 162 | 68 | 30
  Week 192 | -56.3 (17.25) | -52.1 (16.56) | -55.1 (20.69)
  Week 204: number analyzed (Participants) | 158 | 69 | 30
  Week 204 | -58.0 (16.73) | -52.9 (18.09) | -54.7 (19.50)
  Week 216: number analyzed (Participants) | 151 | 63 | 31
  Week 216 | -58.3 (16.50) | -50.8 (18.27) | -51.3 (20.42)
  Week 228: number analyzed (Participants) | 146 | 55 | 30
  Week 228 | -56.3 (19.63) | -53.2 (17.28) | -55.0 (19.69)
  Week 240: number analyzed (Participants) | 148 | 61 | 29
  Week 240 | -58.1 (17.63) | -52.8 (16.04) | -49.6 (18.67)
  Week 252: number analyzed (Participants) | 141 | 55 | 31
  Week 252 | -57.2 (17.56) | -53.9 (17.10) | -52.2 (18.12)
  Week 264: number analyzed (Participants) | 130 | 52 | 29
  Week 264 | -56.5 (16.68) | -50.4 (18.09) | -46.4 (18.60)
  Week 276: number analyzed (Participants) | 123 | 52 | 28
  Week 276 | -56.9 (16.79) | -53.5 (17.07) | -50.1 (17.96)
  Week 288: number analyzed (Participants) | 132 | 51 | 29
  Week 288 | -57.3 (18.97) | -56.3 (17.25) | -49.4 (16.31)
  Week 300: number analyzed (Participants) | 126 | 50 | 25
  Week 300 | -56.8 (17.93) | -52.9 (17.33) | -53.6 (17.36)
  Week 312: number analyzed (Participants) | 125 | 45 | 26
  Week 312 | -58.7 (16.12) | -55.2 (17.19) | -49.4 (17.96)

17. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity Over Time
Description: The participant was asked to rate their current RA disease activity over the past 24 hours on a 100 mm VAS, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity.
Time Frame: as for outcome 1
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 305 | 146 | 37
score on a scale
  Week 6: number analyzed (Participants) | 280 | 145 | 36
  Week 6 | -35.4 (29.83) | -27.2 (27.74) | -26.1 (27.46)
  Week 12: number analyzed (Participants) | 275 | 143 | 36
  Week 12 | -37.5 (29.00) | -29.2 (28.05) | -31.3 (23.13)
  Week 24: number analyzed (Participants) | 257 | 132 | 36
  Week 24 | -36.9 (28.97) | -30.4 (31.16) | -32.9 (25.63)
  Week 36: number analyzed (Participants) | 246 | 126 | 35
  Week 36 | -37.1 (30.36) | -32.6 (28.62) | -34.9 (26.00)
  Week 48: number analyzed (Participants) | 229 | 116 | 36
  Week 48 | -39.2 (30.36) | -30.7 (30.46) | -23.6 (26.58)
  Week 60: number analyzed (Participants) | 219 | 110 | 35
  Week 60 | -40.8 (28.95) | -34.4 (28.36) | -38.3 (24.46)
  Week 72: number analyzed (Participants) | 208 | 104 | 33
  Week 72 | -40.3 (27.36) | -32.1 (30.19) | -26.3 (30.70)
  Week 84: number analyzed (Participants) | 209 | 99 | 33
  Week 84 | -40.1 (30.37) | -32.0 (31.27) | -39.4 (21.35)
  Week 96: number analyzed (Participants) | 205 | 96 | 33
  Week 96 | -38.1 (30.34) | -33.5 (33.51) | -33.5 (22.08)
  Week 108: number analyzed (Participants) | 195 | 93 | 33
  Week 108 | -40.8 (29.75) | -35.0 (29.93) | -32.1 (20.65)
  Week 120: number analyzed (Participants) | 188 | 87 | 30
  Week 120 | -40.6 (29.76) | -32.4 (32.91) | -36.6 (28.02)
  Week 132: number analyzed (Participants) | 184 | 82 | 30
  Week 132 | -40.1 (29.99) | -37.0 (28.43) | -38.4 (27.02)
  Week 144: number analyzed (Participants) | 183 | 75 | 28
  Week 144 | -37.7 (30.73) | -36.8 (28.24) | -33.9 (29.68)
  Week 156: number analyzed (Participants) | 180 | 74 | 28
  Week 156 | -39.7 (32.65) | -36.9 (25.93) | -38.6 (21.61)
  Week 168: number analyzed (Participants) | 177 | 73 | 29
  Week 168 | -42.7 (29.04) | -37.9 (29.10) | -39.0 (32.84)
  Week 180: number analyzed (Participants) | 179 | 71 | 29
  Week 180 | -40.3 (29.52) | -30.7 (33.34) | -33.3 (34.03)
  Week 192: number analyzed (Participants) | 170 | 72 | 30
  Week 192 | -41.0 (28.73) | -33.4 (33.30) | -42.1 (23.97)
  Week 204: number analyzed (Participants) | 166 | 71 | 30
  Week 204 | -42.0 (29.28) | -33.2 (34.00) | -43.7 (25.60)
  Week 216: number analyzed (Participants) | 161 | 65 | 30
  Week 216 | -39.0 (32.18) | -32.5 (30.72) | -35.6 (27.03)
  Week 228: number analyzed (Participants) | 153 | 59 | 30
  Week 228 | -38.4 (32.29) | -28.5 (37.86) | -40.1 (24.11)
  Week 240: number analyzed (Participants) | 155 | 62 | 28
  Week 240 | -41.9 (30.43) | -37.6 (28.56) | -33.3 (29.03)
  Week 252: number analyzed (Participants) | 151 | 59 | 30
  Week 252 | -40.6 (32.12) | -33.8 (31.76) | -33.5 (35.96)
  Week 264: number analyzed (Participants) | 140 | 55 | 28
  Week 264 | -38.5 (31.53) | -31.6 (34.26) | -32.7 (34.87)
  Week 276: number analyzed (Participants) | 130 | 54 | 27
  Week 276 | -42.4 (27.53) | -36.8 (29.40) | -26.0 (33.79)
  Week 288: number analyzed (Participants) | 138 | 53 | 28
  Week 288 | -43.3 (27.99) | -38.5 (32.21) | -32.2 (28.16)
  Week 300: number analyzed (Participants) | 134 | 52 | 27
  Week 300 | -38.8 (29.04) | -33.4 (34.89) | -31.6 (25.93)
  Week 312: number analyzed (Participants) | 137 | 49 | 27
  Week 312 | -36.5 (32.10) | -39.4 (30.60) | -37.7 (29.67)

18. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain Over Time
Description: Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale from 0 to 100 mm. A score of 0 mm indicates "no pain" and a score of 100 mm indicates "worst possible pain."
Time Frame: as for outcome 1
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 305 | 146 | 37
score on a scale
  Week 6: number analyzed (Participants) | 280 | 145 | 36
  Week 6 | -38.5 (27.16) | -29.9 (24.46) | -30.0 (26.37)
  Week 12: number analyzed (Participants) | 275 | 143 | 36
  Week 12 | -41.3 (26.07) | -29.9 (26.20) | -31.9 (20.23)
  Week 24: number analyzed (Participants) | 257 | 132 | 36
  Week 24 | -42.2 (25.41) | -30.9 (28.77) | -36.0 (21.73)
  Week 36: number analyzed (Participants) | 246 | 126 | 35
  Week 36 | -40.6 (26.41) | -34.6 (26.56) | -34.8 (21.83)
  Week 48: number analyzed (Participants) | 229 | 116 | 36
  Week 48 | -42.4 (26.50) | -31.9 (28.73) | -32.6 (23.67)
  Week 60: number analyzed (Participants) | 219 | 110 | 35
  Week 60 | -41.9 (27.89) | -32.2 (26.50) | -38.6 (23.34)
  Week 72: number analyzed (Participants) | 208 | 104 | 33
  Week 72 | -42.5 (24.76) | -32.0 (25.38) | -31.4 (22.95)
  Week 84: number analyzed (Participants) | 209 | 99 | 33
  Week 84 | -42.1 (25.87) | -33.3 (26.52) | -43.0 (20.51)
  Week 96: number analyzed (Participants) | 205 | 96 | 33
  Week 96 | -40.5 (28.02) | -34.2 (26.14) | -37.6 (20.15)
  Week 108: number analyzed (Participants) | 195 | 93 | 33
  Week 108 | -43.6 (26.28) | -33.9 (27.60) | -36.3 (23.12)
  Week 120: number analyzed (Participants) | 188 | 87 | 30
  Week 120 | -43.0 (26.67) | -36.2 (27.69) | -41.9 (21.40)
  Week 132: number analyzed (Participants) | 184 | 82 | 30
  Week 132 | -42.2 (26.89) | -36.7 (26.71) | -34.4 (27.27)
  Week 144: number analyzed (Participants) | 183 | 75 | 28
  Week 144 | -41.7 (27.02) | -36.7 (27.14) | -33.8 (24.60)
  Week 156: number analyzed (Participants) | 180 | 74 | 28
  Week 156 | -43.5 (25.72) | -37.4 (25.27) | -34.6 (24.91)
  Week 168: number analyzed (Participants) | 177 | 73 | 29
  Week 168 | -43.6 (27.19) | -38.8 (27.67) | -41.6 (25.76)
  Week 180: number analyzed (Participants) | 179 | 71 | 29
  Week 180 | -42.7 (26.54) | -33.6 (30.24) | -36.5 (29.20)
  Week 192: number analyzed (Participants) | 170 | 72 | 30
  Week 192 | -41.6 (27.90) | -33.8 (29.13) | -39.9 (25.44)
  Week 204: number analyzed (Participants) | 166 | 71 | 30
  Week 204 | -44.4 (25.26) | -33.4 (33.05) | -41.9 (22.39)
  Week 216: number analyzed (Participants) | 161 | 65 | 30
  Week 216 | -42.2 (28.01) | -32.5 (32.06) | -33.6 (25.98)
  Week 228: number analyzed (Participants) | 153 | 59 | 30
  Week 228 | -45.1 (24.96) | -29.6 (35.17) | -39.8 (24.70)
  Week 240: number analyzed (Participants) | 155 | 62 | 28
  Week 240 | -43.4 (27.78) | -34.1 (31.98) | -36.1 (25.38)
  Week 252: number analyzed (Participants) | 151 | 59 | 30
  Week 252 | -44.4 (27.49) | -34.3 (28.12) | -38.3 (24.92)
  Week 264: number analyzed (Participants) | 140 | 55 | 28
  Week 264 | -44.0 (25.43) | -35.6 (31.33) | -38.2 (24.11)
  Week 276: number analyzed (Participants) | 130 | 54 | 27
  Week 276 | -46.3 (24.53) | -35.6 (27.39) | -34.1 (26.80)
  Week 288: number analyzed (Participants) | 138 | 53 | 28
  Week 288 | -46.2 (25.61) | -37.6 (28.74) | -33.3 (23.30)
  Week 300: number analyzed (Participants) | 134 | 52 | 27
  Week 300 | -43.0 (25.18) | -34.7 (32.36) | -29.9 (30.21)
  Week 312: number analyzed (Participants) | 137 | 49 | 27
  Week 312 | -44.1 (25.87) | -40.3 (27.37) | -33.4 (30.11)

19. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Over Time
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
Time Frame: as for outcome 1
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 304 | 146 | 37
score on a scale
  Week 6: number analyzed (Participants) | 264 | 136 | 35
  Week 6 | -0.7 (0.62) | -0.6 (0.56) | -0.6 (0.47)
  Week 12: number analyzed (Participants) | 264 | 138 | 34
  Week 12 | -0.7 (0.64) | -0.6 (0.63) | -0.7 (0.55)
  Week 24: number analyzed (Participants) | 236 | 130 | 33
  Week 24 | -0.8 (0.60) | -0.6 (0.61) | -0.7 (0.58)
  Week 36: number analyzed (Participants) | 235 | 117 | 32
  Week 36 | -0.7 (0.66) | -0.6 (0.62) | -0.7 (0.66)
  Week 48: number analyzed (Participants) | 213 | 111 | 34
  Week 48 | -0.8 (0.63) | -0.7 (0.61) | -0.7 (0.58)
  Week 60: number analyzed (Participants) | 206 | 104 | 34
  Week 60 | -0.8 (0.67) | -0.7 (0.66) | -0.7 (0.52)
  Week 72: number analyzed (Participants) | 194 | 100 | 33
  Week 72 | -0.8 (0.65) | -0.7 (0.63) | -0.7 (0.54)
  Week 84: number analyzed (Participants) | 196 | 90 | 32
  Week 84 | -0.9 (0.62) | -0.7 (0.64) | -0.7 (0.57)
  Week 96: number analyzed (Participants) | 192 | 89 | 30
  Week 96 | -0.8 (0.64) | -0.8 (0.69) | -0.8 (0.52)
  Week 108: number analyzed (Participants) | 185 | 87 | 33
  Week 108 | -0.9 (0.67) | -0.7 (0.67) | -0.7 (0.58)
  Week 120: number analyzed (Participants) | 178 | 84 | 29
  Week 120 | -0.8 (0.64) | -0.7 (0.64) | -0.8 (0.62)
  Week 132: number analyzed (Participants) | 176 | 75 | 28
  Week 132 | -0.9 (0.66) | -0.7 (0.64) | -0.8 (0.51)
  Week 144: number analyzed (Participants) | 170 | 70 | 27
  Week 144 | -0.8 (0.72) | -0.8 (0.68) | -0.7 (0.61)
  Week 156: number analyzed (Participants) | 172 | 72 | 26
  Week 156 | -0.8 (0.69) | -0.7 (0.57) | -0.8 (0.61)
  Week 168: number analyzed (Participants) | 168 | 72 | 27
  Week 168 | -0.8 (0.68) | -0.7 (0.67) | -0.8 (0.60)
  Week 180: number analyzed (Participants) | 169 | 69 | 28
  Week 180 | -0.8 (0.70) | -0.7 (0.70) | -0.7 (0.64)
  Week 192: number analyzed (Participants) | 160 | 66 | 26
  Week 192 | -0.8 (0.68) | -0.7 (0.69) | -0.8 (0.57)
  Week 204: number analyzed (Participants) | 160 | 69 | 28
  Week 204 | -0.9 (0.68) | -0.7 (0.79) | -0.8 (0.51)
  Week 216: number analyzed (Participants) | 155 | 64 | 30
  Week 216 | -0.8 (0.69) | -0.7 (0.73) | -0.8 (0.61)
  Week 228: number analyzed (Participants) | 146 | 57 | 29
  Week 228 | -0.9 (0.72) | -0.7 (0.77) | -0.7 (0.61)
  Week 240: number analyzed (Participants) | 146 | 62 | 28
  Week 240 | -0.8 (0.69) | -0.7 (0.77) | -0.6 (0.61)
  Week 252: number analyzed (Participants) | 139 | 57 | 27
  Week 252 | -0.9 (0.69) | -0.7 (0.77) | -0.7 (0.59)
  Week 264: number analyzed (Participants) | 136 | 50 | 27
  Week 264 | -0.8 (0.68) | -0.7 (0.65) | -0.7 (0.59)
  Week 276: number analyzed (Participants) | 127 | 52 | 27
  Week 276 | -0.8 (0.69) | -0.6 (0.66) | -0.7 (0.61)
  Week 288: number analyzed (Participants) | 125 | 47 | 26
  Week 288 | -0.9 (0.70) | -0.7 (0.74) | -0.8 (0.61)
  Week 300: number analyzed (Participants) | 128 | 51 | 24
  Week 300 | -0.8 (0.76) | -0.7 (0.70) | -0.7 (0.68)
  Week 312: number analyzed (Participants) | 129 | 46 | 27
  Week 312 | -0.8 (0.71) | -0.8 (0.74) | -0.7 (0.69)

20. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP) Over Time
Time Frame: as for outcome 1
Population: Open-label treated population with available data at each time point
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 306 | 149 | 38
mg/L
  Week 6: number analyzed (Participants) | 297 | 149 | 38
  Week 6 | -7.9 (21.74) | -10.0 (21.95) | -13.0 (29.00)
  Week 12: number analyzed (Participants) | 282 | 147 | 38
  Week 12 | -9.0 (18.96) | -10.7 (20.94) | -12.8 (26.93)
  Week 24: number analyzed (Participants) | 264 | 139 | 38
  Week 24 | -9.4 (17.38) | -7.2 (36.97) | -9.1 (29.38)
  Week 36: number analyzed (Participants) | 254 | 133 | 38
  Week 36 | -9.5 (18.62) | -11.1 (22.03) | -13.5 (28.34)
  Week 48: number analyzed (Participants) | 239 | 125 | 38
  Week 48 | -8.8 (17.50) | -10.2 (22.28) | -13.3 (22.69)
  Week 60: number analyzed (Participants) | 227 | 117 | 37
  Week 60 | -9.6 (17.78) | -10.3 (22.10) | -11.0 (21.62)
  Week 72: number analyzed (Participants) | 222 | 111 | 36
  Week 72 | -9.2 (19.42) | -9.9 (22.95) | -11.2 (20.16)
  Week 84: number analyzed (Participants) | 217 | 105 | 35
  Week 84 | -8.3 (24.66) | -10.0 (28.56) | -10.2 (16.57)
  Week 96: number analyzed (Participants) | 213 | 101 | 35
  Week 96 | -10.1 (17.74) | -10.3 (22.36) | -11.1 (17.61)
  Week 108: number analyzed (Participants) | 206 | 96 | 35
  Week 108 | -9.8 (21.56) | -10.7 (19.36) | -10.8 (17.39)
  Week 120: number analyzed (Participants) | 198 | 91 | 32
  Week 120 | -8.4 (18.27) | -10.9 (19.63) | -9.2 (18.62)
  Week 132: number analyzed (Participants) | 181 | 83 | 33
  Week 132 | -8.9 (15.19) | -9.0 (21.32) | -9.3 (17.53)
  Week 144: number analyzed (Participants) | 180 | 76 | 32
  Week 144 | -7.3 (17.15) | -9.9 (23.45) | -5.9 (26.82)
  Week 156: number analyzed (Participants) | 176 | 72 | 32
  Week 156 | -8.6 (16.60) | -6.0 (52.17) | -10.9 (18.20)
  Week 168: number analyzed (Participants) | 171 | 74 | 32
  Week 168 | -7.7 (18.37) | -7.5 (28.96) | -8.8 (17.88)
  Week 180: number analyzed (Participants) | 185 | 72 | 32
  Week 180 | -10.0 (19.41) | -10.3 (21.44) | -9.2 (19.16)
  Week 192: number analyzed (Participants) | 177 | 73 | 30
  Week 192 | -9.4 (23.81) | -9.9 (21.04) | -9.3 (20.07)
  Week 204: number analyzed (Participants) | 174 | 72 | 32
  Week 204 | -8.4 (28.90) | -9.6 (21.29) | -9.0 (19.07)
  Week 216: number analyzed (Participants) | 166 | 68 | 32
  Week 216 | -11.5 (20.22) | -10.0 (22.42) | -8.4 (19.70)
  Week 228: number analyzed (Participants) | 165 | 61 | 31
  Week 228 | -11.0 (20.71) | -12.2 (20.89) | -10.0 (17.46)
  Week 240: number analyzed (Participants) | 163 | 63 | 32
  Week 240 | -10.6 (24.45) | -9.1 (22.38) | -9.2 (17.55)
  Week 252: number analyzed (Participants) | 151 | 61 | 31
  Week 252 | -10.4 (19.33) | -9.4 (24.28) | -9.9 (18.83)
  Week 264: number analyzed (Participants) | 141 | 57 | 28
  Week 264 | -11.2 (21.02) | -9.9 (23.99) | -11.1 (18.19)
  Week 276: number analyzed (Participants) | 135 | 56 | 27
  Week 276 | -10.5 (18.04) | -11.2 (20.20) | -10.9 (17.95)
  Week 288: number analyzed (Participants) | 115 | 51 | 26
  Week 288 | -10.6 (16.09) | -12.9 (21.85) | -7.5 (14.48)
  Week 300: number analyzed (Participants) | 113 | 40 | 22
  Week 300 | -11.1 (14.63) | -11.4 (21.67) | -11.0 (19.69)
  Week 312: number analyzed (Participants) | 124 | 49 | 29
  Week 312 | -10.3 (22.22) | -12.0 (21.14) | -8.7 (15.19)

21. Secondary Outcome: Change From Baseline in in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale Over Time
Description: The FACIT Fatigue scale is a 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past 7 days. Each of the fatigue and impact of fatigue items are measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The FACIT Fatigue Scale is the sum of the individual 13 scores and ranges from 0 to 52 where higher scores indicate better quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline (of the preceding RCT study) and Weeks 6, 12, 24, 36, 48, 72, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, and 312
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 304 | 146 | 37
score on a scale
  Week 6: number analyzed (Participants) | 278 | 145 | 36
  Week 6 | 9.5 (10.50) | 9.0 (9.69) | 8.8 (9.26)
  Week 12: number analyzed (Participants) | 275 | 142 | 36
  Week 12 | 9.9 (10.49) | 8.7 (10.87) | 8.6 (10.43)
  Week 24: number analyzed (Participants) | 256 | 133 | 36
  Week 24 | 10.7 (10.04) | 10.6 (11.60) | 8.3 (9.65)
  Week 36: number analyzed (Participants) | 244 | 126 | 35
  Week 36 | 10.1 (10.59) | 10.0 (11.58) | 8.0 (11.50)
  Week 48: number analyzed (Participants) | 228 | 116 | 36
  Week 48 | 10.4 (10.58) | 10.8 (10.44) | 8.4 (10.83)
  Week 72: number analyzed (Participants) | 208 | 107 | 33
  Week 72 | 10.8 (9.55) | 10.9 (10.64) | 9.2 (11.44)
  Week 96: number analyzed (Participants) | 204 | 96 | 32
  Week 96 | 10.3 (10.45) | 11.7 (12.72) | 9.5 (11.27)
  Week 108: number analyzed (Participants) | 194 | 93 | 33
  Week 108 | 10.5 (10.49) | 11.9 (12.08) | 7.9 (10.62)
  Week 120: number analyzed (Participants) | 187 | 87 | 30
  Week 120 | 11.0 (10.76) | 11.6 (11.95) | 10.7 (11.30)
  Week 132: number analyzed (Participants) | 182 | 82 | 30
  Week 132 | 11.4 (10.13) | 10.7 (11.47) | 10.7 (10.36)
  Week 144: number analyzed (Participants) | 182 | 75 | 28
  Week 144 | 9.9 (11.36) | 11.2 (12.09) | 9.8 (11.67)
  Week 156: number analyzed (Participants) | 179 | 74 | 28
  Week 156 | 10.6 (10.94) | 11.2 (11.48) | 8.6 (12.32)
  Week 168: number analyzed (Participants) | 176 | 73 | 29
  Week 168 | 10.8 (12.27) | 10.6 (12.46) | 11.4 (13.18)
  Week 180: number analyzed (Participants) | 178 | 71 | 29
  Week 180 | 11.0 (11.59) | 9.6 (13.56) | 11.4 (12.45)
  Week 192: number analyzed (Participants) | 169 | 72 | 30
  Week 192 | 10.8 (10.50) | 10.9 (11.82) | 11.5 (13.27)
  Week 204: number analyzed (Participants) | 164 | 71 | 30
  Week 204 | 11.3 (10.56) | 10.2 (13.01) | 11.2 (12.70)
  Week 216: number analyzed (Participants) | 160 | 65 | 30
  Week 216 | 11.4 (11.93) | 10.4 (13.92) | 10.1 (12.87)
  Week 228: number analyzed (Participants) | 152 | 59 | 30
  Week 228 | 11.0 (11.25) | 10.8 (14.00) | 11.1 (13.18)
  Week 240: number analyzed (Participants) | 154 | 62 | 28
  Week 240 | 11.9 (10.93) | 11.4 (13.08) | 9.2 (13.81)
  Week 252: number analyzed (Participants) | 150 | 59 | 30
  Week 252 | 11.5 (10.83) | 10.2 (13.68) | 8.4 (13.48)
  Week 264: number analyzed (Participants) | 139 | 55 | 28
  Week 264 | 11.6 (10.95) | 10.7 (12.52) | 7.8 (13.94)
  Week 276: number analyzed (Participants) | 129 | 54 | 27
  Week 276 | 12.1 (10.98) | 9.2 (13.02) | 7.3 (13.02)
  Week 288: number analyzed (Participants) | 137 | 53 | 28
  Week 288 | 11.6 (10.88) | 12.3 (11.83) | 9.0 (13.94)
  Week 300: number analyzed (Participants) | 133 | 52 | 27
  Week 300 | 11.1 (11.14) | 9.7 (13.12) | 7.0 (13.46)
  Week 312: number analyzed (Participants) | 136 | 49 | 27
  Week 312 | 10.7 (11.24) | 11.6 (12.67) | 8.6 (14.35)

22. Secondary Outcome: Change From Baseline in Work Instability Scale for RA (RA-WIS) Over Time
Description: RA-WIS is a tool to evaluate work instability (the consequence of a mismatch between an individual's functional ability and their work tasks). RA-WIS consists of 23 questions relating to the participant's functioning in their work environment, each answered as Yes or No. The total score is the number of questions answered Yes, and ranges from 0 to 23.
  A score < 10 means low risk, scores between 10 and 17 indicate medium risk, and scores > 17 indicate high risk of work instability.
  A negative change from Baseline indicates improvement in work instability.
Time Frame: as for outcome 21
Population: Open-label treated population who were currently working at Baseline and at each visit visit and with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 87 | 53 | 13
score on a scale
  Week 6: number analyzed (Participants) | 75 | 45 | 12
  Week 6 | -6.2 (5.55) | -3.3 (5.51) | -4.1 (3.00)
  Week 12: number analyzed (Participants) | 70 | 43 | 12
  Week 12 | -6.6 (6.16) | -4.0 (6.32) | -4.2 (3.35)
  Week 24: number analyzed (Participants) | 67 | 41 | 12
  Week 24 | -7.0 (6.51) | -4.6 (6.63) | -3.6 (3.53)
  Week 36: number analyzed (Participants) | 61 | 42 | 11
  Week 36 | -6.8 (6.29) | -4.6 (6.21) | -3.3 (6.18)
  Week 48: number analyzed (Participants) | 55 | 40 | 12
  Week 48 | -6.8 (5.94) | -5.0 (6.47) | -3.5 (4.98)
  Week 72: number analyzed (Participants) | 51 | 39 | 12
  Week 72 | -7.5 (6.83) | -4.8 (6.27) | -4.3 (4.10)
  Week 96: number analyzed (Participants) | 54 | 37 | 12
  Week 96 | -6.5 (6.72) | -6.3 (7.55) | -4.0 (4.18)
  Week 108: number analyzed (Participants) | 52 | 32 | 11
  Week 108 | -6.8 (6.80) | -6.5 (6.71) | -3.5 (4.80)
  Week 120: number analyzed (Participants) | 47 | 31 | 9
  Week 120 | -7.6 (6.66) | -5.1 (7.38) | -5.7 (4.44)
  Week 132: number analyzed (Participants) | 47 | 29 | 10
  Week 132 | -7.2 (6.04) | -5.6 (6.99) | -4.7 (3.47)
  Week 144: number analyzed (Participants) | 46 | 26 | 8
  Week 144 | -5.9 (6.51) | -5.6 (7.65) | -4.3 (3.41)
  Week 156: number analyzed (Participants) | 47 | 25 | 8
  Week 156 | -6.2 (7.13) | -4.3 (7.62) | -4.9 (3.72)
  Week 168: number analyzed (Participants) | 43 | 24 | 8
  Week 168 | -5.8 (6.01) | -4.3 (6.96) | -5.1 (6.69)
  Week 180: number analyzed (Participants) | 43 | 24 | 6
  Week 180 | -5.3 (6.61) | -3.5 (7.03) | -4.2 (3.19)
  Week 192: number analyzed (Participants) | 40 | 24 | 7
  Week 192 | -5.5 (6.42) | -3.5 (7.36) | -4.3 (2.93)
  Week 204: number analyzed (Participants) | 36 | 23 | 8
  Week 204 | -6.4 (7.06) | -3.7 (7.52) | -5.0 (3.78)
  Week 216: number analyzed (Participants) | 38 | 23 | 9
  Week 216 | -6.0 (7.55) | -3.4 (7.11) | -5.0 (2.92)
  Week 228: number analyzed (Participants) | 38 | 18 | 7
  Week 228 | -6.5 (7.16) | -1.9 (7.55) | -4.6 (4.24)
  Week 240: number analyzed (Participants) | 34 | 21 | 6
  Week 240 | -5.9 (7.05) | -3.1 (7.61) | -4.5 (4.09)
  Week 252: number analyzed (Participants) | 33 | 18 | 8
  Week 252 | -5.8 (6.43) | -2.0 (8.05) | -5.0 (3.70)
  Week 264: number analyzed (Participants) | 33 | 20 | 8
  Week 264 | -5.0 (6.53) | -3.4 (8.00) | -4.5 (3.89)
  Week 276: number analyzed (Participants) | 30 | 18 | 7
  Week 276 | -5.0 (6.74) | -2.7 (8.27) | -5.0 (2.52)
  Week 288: number analyzed (Participants) | 29 | 17 | 8
  Week 288 | -5.0 (7.05) | -4.8 (7.38) | -4.8 (3.45)
  Week 300: number analyzed (Participants) | 30 | 15 | 8
  Week 300 | -4.6 (7.23) | -4.3 (8.51) | -4.6 (4.07)
  Week 312: number analyzed (Participants) | 31 | 15 | 8
  Week 312 | -4.2 (7.00) | -3.9 (8.37) | -2.9 (4.45)

23. Secondary Outcome: Change From Baseline in EuroQoL-5D (EQ-5D) Index Over Time
Description: The EQ-5D-5L is a generic measure of health status consisting of two parts. The first part (the descriptive system) assesses health in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which is rated on 5 levels of severity (1: no problem, 2: slight problems, 3: moderate problems, 4: severe problems, 5: extreme problems).
  A health state index score was calculated from individual health profiles using a UK scoring algorithm. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The higher the score the better the health status. A positive change from baseline indicates improvement in health status.
Time Frame: as for outcome 21
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 304 | 146 | 37
score on a scale
  Week 6: number analyzed (Participants) | 278 | 145 | 36
  Week 6 | 0.2 (0.24) | 0.2 (0.27) | 0.2 (0.18)
  Week 12: number analyzed (Participants) | 275 | 142 | 36
  Week 12 | 0.2 (0.23) | 0.2 (0.29) | 0.2 (0.14)
  Week 24: number analyzed (Participants) | 256 | 133 | 36
  Week 24 | 0.2 (0.23) | 0.2 (0.28) | 0.2 (0.16)
  Week 36: number analyzed (Participants) | 244 | 126 | 35
  Week 36 | 0.2 (0.24) | 0.2 (0.27) | 0.2 (0.16)
  Week 48: number analyzed (Participants) | 228 | 116 | 36
  Week 48 | 0.2 (0.25) | 0.2 (0.31) | 0.1 (0.20)
  Week 72: number analyzed (Participants) | 209 | 107 | 33
  Week 72 | 0.2 (0.24) | 0.2 (0.28) | 0.2 (0.16)
  Week 96: number analyzed (Participants) | 204 | 97 | 32
  Week 96 | 0.2 (0.25) | 0.2 (0.28) | 0.2 (0.15)
  Week 108: number analyzed (Participants) | 194 | 93 | 33
  Week 108 | 0.2 (0.26) | 0.2 (0.28) | 0.1 (0.16)
  Week 120: number analyzed (Participants) | 187 | 87 | 30
  Week 120 | 0.2 (0.26) | 0.2 (0.27) | 0.2 (0.16)
  Week 132: number analyzed (Participants) | 182 | 82 | 30
  Week 132 | 0.2 (0.25) | 0.2 (0.26) | 0.2 (0.15)
  Week 144: number analyzed (Participants) | 182 | 75 | 28
  Week 144 | 0.2 (0.28) | 0.2 (0.27) | 0.2 (0.17)
  Week 156: number analyzed (Participants) | 179 | 74 | 28
  Week 156 | 0.2 (0.27) | 0.2 (0.26) | 0.1 (0.18)
  Week 168: number analyzed (Participants) | 176 | 73 | 29
  Week 168 | 0.2 (0.29) | 0.2 (0.28) | 0.2 (0.20)
  Week 180: number analyzed (Participants) | 178 | 71 | 29
  Week 180 | 0.2 (0.27) | 0.2 (0.33) | 0.2 (0.20)
  Week 192: number analyzed (Participants) | 169 | 72 | 30
  Week 192 | 0.2 (0.27) | 0.2 (0.27) | 0.2 (0.20)
  Week 204: number analyzed (Participants) | 164 | 71 | 30
  Week 204 | 0.2 (0.27) | 0.2 (0.31) | 0.2 (0.21)
  Week 216: number analyzed (Participants) | 160 | 65 | 30
  Week 216 | 0.2 (0.29) | 0.2 (0.30) | 0.2 (0.18)
  Week 228: number analyzed (Participants) | 152 | 59 | 30
  Week 228 | 0.2 (0.26) | 0.2 (0.31) | 0.1 (0.22)
  Week 240: number analyzed (Participants) | 154 | 62 | 28
  Week 240 | 0.3 (0.29) | 0.2 (0.26) | 0.1 (0.22)
  Week 252: number analyzed (Participants) | 150 | 59 | 30
  Week 252 | 0.2 (0.26) | 0.2 (0.28) | 0.2 (0.22)
  Week 264: number analyzed (Participants) | 139 | 55 | 28
  Week 264 | 0.3 (0.29) | 0.2 (0.25) | 0.1 (0.23)
  Week 276: number analyzed (Participants) | 129 | 54 | 27
  Week 276 | 0.2 (0.30) | 0.2 (0.26) | 0.1 (0.22)
  Week 288: number analyzed (Participants) | 137 | 53 | 28
  Week 288 | 0.3 (0.27) | 0.2 (0.27) | 0.1 (0.23)
  Week 300: number analyzed (Participants) | 133 | 52 | 27
  Week 300 | 0.2 (0.28) | 0.2 (0.27) | 0.1 (0.19)
  Week 312: number analyzed (Participants) | 136 | 49 | 27
  Week 312 | 0.2 (0.29) | 0.2 (0.26) | 0.1 (0.25)

24. Secondary Outcome: Change From Baseline in EuroQoL-5D VAS Score Over Time
Description: The EQ-5D-5L is a generic measure of health status consisting of two parts. The second part of the questionnaire consists of a visual analog scale (VAS) on which the participant rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
  A positive change from baseline indicates improvement.
Time Frame: as for outcome 21
Population: Open-label treated population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upadacitinib Never Titrated | Upadacitinib Titrated Up and Not Down | Upadacitinib Titrated Up and Down
Number analyzed (Participants) | 304 | 146 | 37
score on a scale
  Week 6: number analyzed (Participants) | 278 | 145 | 36
  Week 6 | 23.7 (25.21) | 14.4 (24.94) | 21.6 (20.49)
  Week 12: number analyzed (Participants) | 275 | 142 | 36
  Week 12 | 26.0 (25.62) | 15.9 (25.83) | 19.4 (25.07)
  Week 24: number analyzed (Participants) | 256 | 133 | 36
  Week 24 | 27.5 (25.24) | 16.8 (27.31) | 20.7 (20.67)
  Week 36: number analyzed (Participants) | 244 | 126 | 35
  Week 36 | 27.0 (26.29) | 18.6 (27.10) | 18.6 (21.05)
  Week 48: number analyzed (Participants) | 228 | 116 | 36
  Week 48 | 25.9 (26.87) | 19.1 (28.61) | 19.7 (21.07)
  Week 72: number analyzed (Participants) | 209 | 107 | 33
  Week 72 | 28.0 (24.36) | 21.9 (26.33) | 26.7 (21.43)
  Week 96: number analyzed (Participants) | 204 | 97 | 32
  Week 96 | 27.5 (26.86) | 22.4 (27.73) | 25.4 (19.25)
  Week 108: number analyzed (Participants) | 194 | 93 | 33
  Week 108 | 28.8 (25.72) | 23.2 (25.81) | 20.5 (19.06)
  Week 120: number analyzed (Participants) | 187 | 87 | 30
  Week 120 | 28.4 (27.22) | 23.7 (25.36) | 27.2 (23.54)
  Week 132: number analyzed (Participants) | 182 | 82 | 30
  Week 132 | 26.3 (28.75) | 23.5 (26.23) | 28.1 (19.62)
  Week 144: number analyzed (Participants) | 182 | 75 | 28
  Week 144 | 28.6 (26.71) | 23.5 (24.29) | 24.7 (25.32)
  Week 156: number analyzed (Participants) | 179 | 74 | 28
  Week 156 | 29.9 (25.48) | 22.5 (24.62) | 22.1 (23.52)
  Week 168: number analyzed (Participants) | 176 | 73 | 29
  Week 168 | 30.3 (25.29) | 22.6 (23.74) | 28.1 (24.06)
  Week 180: number analyzed (Participants) | 178 | 71 | 29
  Week 180 | 30.0 (24.30) | 22.0 (27.24) | 27.0 (21.68)
  Week 192: number analyzed (Participants) | 169 | 72 | 30
  Week 192 | 29.7 (24.65) | 23.6 (26.41) | 30.8 (21.96)
  Week 204: number analyzed (Participants) | 164 | 71 | 30
  Week 204 | 32.0 (24.41) | 23.1 (27.13) | 30.7 (22.99)
  Week 216: number analyzed (Participants) | 160 | 65 | 30
  Week 216 | 30.0 (26.93) | 24.0 (26.40) | 28.0 (21.73)
  Week 228: number analyzed (Participants) | 152 | 59 | 30
  Week 228 | 31.6 (24.92) | 19.7 (26.70) | 29.5 (23.85)
  Week 240: number analyzed (Participants) | 154 | 62 | 28
  Week 240 | 31.3 (26.18) | 21.9 (25.62) | 28.4 (26.55)
  Week 252: number analyzed (Participants) | 150 | 59 | 30
  Week 252 | 31.2 (24.46) | 22.8 (26.74) | 25.6 (23.74)
  Week 264: number analyzed (Participants) | 139 | 55 | 28
  Week 264 | 30.8 (25.30) | 22.2 (23.60) | 21.9 (24.81)
  Week 276: number analyzed (Participants) | 129 | 54 | 27
  Week 276 | 32.4 (23.37) | 20.5 (25.68) | 25.4 (20.62)
  Week 288: number analyzed (Participants) | 137 | 53 | 28
  Week 288 | 32.3 (24.66) | 24.6 (25.54) | 25.3 (22.57)
  Week 300: number analyzed (Participants) | 133 | 52 | 27
  Week 300 | 30.5 (24.39) | 20.4 (27.31) | 23.6 (17.27)
  Week 312: number analyzed (Participants) | 136 | 49 | 27
  Week 312 | 31.2 (25.15) | 25.8 (24.81) | 24.1 (25.18)

25. Secondary Outcome: Percentage of Participants With Satisfactory Humoral Response to PCV-13 12 Weeks After Vaccination
Description: as for outcome 4
Time Frame: Vaccination Baseline and 12 weeks after vaccination
Population: The sub-study full analysis set (FAS) included all participants enrolled in the sub-study who received PCV-13 vaccination and at least 1 dose of upadacitinib 15 mg or 30 mg after vaccination during the sub-study. Analysis includes participants with available data at the Week 12 visit of the sub-study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 15 mg + PCV-13 | Upadacitinib 30 mg + PCV-13
Number analyzed (Participants) | 79 | 22
percentage of participants | 64.6 [54.0 to 75.1] | 54.5 [33.7 to 75.4]

26. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-pneumococcal Antibody Levels to Each of the 12 Pneumococcal Antigens 4 and 12 Weeks After Vaccination
Time Frame: Vaccination Baseline and 4 and 12 weeks after vaccination
Population: Sub-study full analysis set with available data at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Upadacitinib 15 mg + PCV-13 | Upadacitinib 30 mg + PCV-13
Number analyzed (Participants) | 83 | 23
fold-rise
  Antigen 1: Week 4 | 7.90 [6.096 to 10.244] | 6.53 [3.985 to 10.684]
  Antigen 1: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 1: Week 12 | 8.07 [6.158 to 10.567] | 6.54 [3.922 to 10.911]
  Antigen 3: Week 4 | 2.59 [2.088 to 3.205] | 2.30 [1.530 to 3.467]
  Antigen 3: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 3: Week 12 | 2.26 [1.805 to 2.824] | 2.24 [1.464 to 3.431]
  Antigen 4: Week 4 | 5.61 [4.279 to 7.362] | 3.82 [2.283 to 6.402]
  Antigen 4: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 4: Week 12 | 5.17 [3.888 to 6.885] | 3.39 [1.970 to 5.826]
  Antigen 5: Week 4 | 1.90 [1.521 to 2.366] | 1.60 [1.050 to 2.431]
  Antigen 5: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 5: Week 12 | 1.84 [1.485 to 2.288] | 1.57 [1.043 to 2.367]
  Antigen 6B: Week 4 | 4.50 [3.325 to 6.077] | 3.10 [1.748 to 5.511]
  Antigen 6B: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 6B: Week 12 | 3.90 [2.801 to 5.436] | 3.25 [1.732 to 6.092]
  Antigen 7F: Week 4 | 3.58 [2.824 to 4.548] | 2.83 [1.797 to 4.446]
  Antigen 7F: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 7F: Week 12 | 3.30 [2.552 to 4.255] | 3.02 [1.856 to 4.897]
  Antigen 9V: Week 4 | 5.69 [4.260 to 7.611] | 2.76 [1.588 to 4.794]
  Antigen 9V: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 9V: Week 12 | 6.18 [4.583 to 8.325] | 2.91 [1.649 to 5.138]
  Antigen 14: Week 4 | 2.97 [2.373 to 3.723] | 2.42 [1.573 to 3.707]
  Antigen 14: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 14: Week 12 | 2.84 [2.231 to 3.613] | 2.41 [1.524 to 3.804]
  Antigen 18C: Week 4 | 4.52 [3.526 to 5.801] | 3.23 [2.009 to 5.179]
  Antigen 18C: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 18C: Week 12 | 4.42 [3.443 to 5.670] | 3.53 [2.201 to 5.666]
  Antigen 19A: Week 4 | 1.47 [1.264 to 1.702] | 1.12 [0.844 to 1.485]
  Antigen 19A: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 19A: Week 12 | 1.44 [1.245 to 1.666] | 1.15 [0.876 to 1.521]
  Antigen 19F: Week 4 | 2.27 [1.834 to 2.808] | 2.32 [1.549 to 3.476]
  Antigen 19F: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 19F: Week 12 | 2.17 [1.761 to 2.671] | 1.99 [1.344 to 2.958]
  Antigen 23F: Week 4 | 4.32 [3.291 to 5.672] | 3.11 [1.855 to 5.218]
  Antigen 23F: Week 12: number analyzed (Participants) | 79 | 22
  Antigen 23F: Week 12 | 4.06 [3.048 to 5.413] | 3.29 [1.908 to 5.666]

ADVERSE EVENTS:
Time Frame: From the first dose of open-label upadacitinib up to 30 days after the last dose, up to 316 weeks.
Groups:
- Upadacitinib 6 mg BID/15 mg QD: Participants received upadacitinib 6 mg BID. From January 2017 participants were transitioned to 15 mg upadacitinib QD. Includes events that occurred until the time of up-titration for participants who were up-titrated.
- Upadacitinib 12 mg BID/30 mg QD: Participants received upadacitinib 12 mg BID. From January 2017 participants were transitioned to 30 mg upadacitinib QD. Includes events that occurred from the time of up-titration until time of down titration to 6 mg BID/15 mg QD for participants who titrated up and back down.
- Upadacitinib 6 mg BID/15 mg QD Post Down-titration: Participants who down-titrated to 6 mg BID/15 mg QD after up-titration to 15 mg BID/30 mg QD. Includes events that occurred after down titration.
Arm/Group | Upadacitinib 6 mg BID/15 mg QD | Upadacitinib 12 mg BID/30 mg QD | Upadacitinib 6 mg BID/15 mg QD Post Down-titration
All-Cause Mortality (participants affected / at risk) | 5/493 | 3/187 | 0/38
Serious Adverse Events (participants affected / at risk) | 68/493 | 42/187 | 5/38
Other Adverse Events (participants affected / at risk) | 233/493 | 113/187 | 23/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upadacitinib 6 mg BID/15 mg QD (N=493) | Upadacitinib 12 mg BID/30 mg QD (N=187) | Upadacitinib 6 mg BID/15 mg QD Post Down-titration (N=38)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISSECTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
GOITRE (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
CORNEAL PERFORATION (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
MACULAR HOLE (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEATH (General disorders) | 2 (2) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENDOMETRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS A (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
HISTOPLASMOSIS DISSEMINATED (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LATENT TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 7 (7) | 3 (3) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VARICELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
INCARCERATED INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
CLEAR CELL RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
INVASIVE LOBULAR BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
INVASIVE PAPILLARY BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SEBACEOUS CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
THYROID B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BRAIN STEM INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OCCIPITAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DEVICE LOOSENING (Product Issues) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
DISSOCIATIVE DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
BLADDER PROLAPSE (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
HYDROSALPINX (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PARANASAL CYST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upadacitinib 6 mg BID/15 mg QD (N=493) | Upadacitinib 12 mg BID/30 mg QD (N=187) | Upadacitinib 6 mg BID/15 mg QD Post Down-titration (N=38)
ANAEMIA (Blood and lymphatic system disorders) | 7 (7) | 11 (12) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 15 (17) | 5 (6) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 10 (13) | 2 (3) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 7 (7) | 10 (11) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 6 (9) | 10 (11) | 2 (2)
BRONCHITIS (Infections and infestations) | 42 (66) | 14 (23) | 6 (8)
HERPES ZOSTER (Infections and infestations) | 22 (23) | 21 (24) | 3 (3)
LATENT TUBERCULOSIS (Infections and infestations) | 10 (10) | 2 (2) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 3 (4)
NASOPHARYNGITIS (Infections and infestations) | 47 (75) | 16 (19) | 3 (3)
PHARYNGITIS (Infections and infestations) | 10 (12) | 3 (3) | 2 (2)
SINUSITIS (Infections and infestations) | 13 (15) | 14 (24) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 49 (71) | 38 (63) | 3 (8)
URINARY TRACT INFECTION (Infections and infestations) | 47 (84) | 28 (54) | 3 (6)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 7 (8) | 14 (20) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 12 (15) | 4 (4) | 3 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 16 (17) | 5 (5) | 2 (3)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 34 (44) | 17 (27) | 3 (4)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 29 (35) | 17 (18) | 3 (3)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 21 (32) | 21 (35) | 0 (0) — The Preferred Term of rheumatoid arthritis was due to the reported term of "worsening of RA" being coded to rheumatoid arthritis.
HEADACHE (Nervous system disorders) | 18 (23) | 5 (7) | 3 (3)
NEPHROLITHIASIS (Renal and urinary disorders) | 7 (10) | 1 (1) | 2 (3)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 10 (11) | 1 (2)
RASH (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 2 (2)
ROSACEA (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2)
HYPERTENSION (Vascular disorders) | 22 (23) | 19 (19) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02049138/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT02049138/SAP_001.pdf